J1P-MC-KFAH Statistical Analysis Plan Version 1

An Adaptive Phase 2, Randomized, Double-Blind, Placebo-Controlled Study of LY3471851 (NKTR-358) in Patients with Moderately to Severely Active Ulcerative Colitis

NCT04677179

Approval Date: 18 Mar 2022

**Protocol Title:** An Adaptive Phase 2, Randomized, Double-Blind, Placebo-Controlled Study of LY3471851 (NKTR-358) in Patients with Moderately to Severely Active Ulcerative Colitis

**Protocol Number:** J1P-MC-KFAH

Compound Number: LY3471851

**Short Title: INSTRUCT-UC** 

Sponsor Name: Eli Lilly and Company

Legal Registered Address: Indianapolis, Indiana USA 46285

**Regulatory Agency Identifier Number(s)** 

**Registry** ID

IND 151216

EudraCT 2020-003017-35

## **Confidential Information**

The information contained in this document is confidential and the information contained within it may not be reproduced or otherwise disseminated without the approval of Eli Lilly and Company or its subsidiaries

**Note to Regulatory Authorities**: This document may contain protected personal data and/or commercially confidential information exempt from public disclosure. Eli Lilly and Company requests consultation regarding release/redaction prior to any public release. In the United States, this document is subject to Freedom of Information Act (FOIA) Exemption 4 and may not be reproduced or otherwise disseminated without the written approval of Eli Lilly and Company or its subsidiaries.

## **Table of Contents**

| Table ( | of Contents | 2 |
|---|---|---|
| Versio | n history | 4 |
| 1. | Introduction | 5 |
| 1.1. | Objectives, Endpoints, and Estimands | |
| 1.2. | Study Design | |
| 1.2.1. | Method of Assignment to Treatment | |
| 2. | Statistical Hypotheses | |
| 2.1. | Multiplicity Adjustment. | |
| 3. | Analysis Sets | |
| 4. | Statistical Analyses | |
| 4.1. | General Considerations. | |
| 4.1.1. | Analysis Methods. | |
| 4.1.2. | Handling of Dropouts or Missing Data | |
| 4.2. | Participant Dispositions | |
| 4.3. | Primary Endpoint Analysis | |
| 4.3.1. | Definition of endpoint. | |
| 4.3.2. | Main analytical approach | |
| 4.3.3. | Bayesian Model Averaging. | |
| 4.4. | Secondary Endpoints Analyses | |
| 4.4.1. | Secondary Efficacy Endpoints | |
| 4.4.2. | Secondary Health Outcome Endpoints | |
| 4.4.3. | Bioanalytical and Pharmacokinetic/Pharmacodynamic Methods | |
| 4.5. | Tertiary/Exploratory Endpoints Analyses | |
| 4.5.1. | Exploratory Efficacy Analysis | 25 |
| 4.6. | Safety Analyses | 26 |
| 4.6.1. | Extent of Exposure | 27 |
| 4.6.2. | Adverse Events | |
| 4.6.3. | Adverse Events of Special Interest | 30 |
| 4.6.4. | Injection Site Reaction | 33 |
| 4.6.5. | Clinical Laboratory Evaluation | 34 |
| 4.6.6. | Vital Signs and Other Physical Characteristics | 37 |
| 4.6.7. | Electrocardiograms | <u></u> 38 |
| 4.6.8. | CCI | 38 |
| 4.7. | Other Analyses | |
| 4.7.1. | Efficacy Subgroup Analysis | |
| 4.7.2. | Safety Subgroup Analyses | |
| 4.8. | Interim Analyses | |
| 4.8.1. | Data Monitoring Committee (DMC) | |
| 4.9. | Changes to Protocol-Planned Analyses | 42 |
| 5. | Sample Size Determination | 43 |
| 6. | Supporting Documentation | |
| 6.1. | Appendix 1: Demographic and Baseline Characteristics | 44 |

## CONFIDENTIAL

| <b>7.</b> | References | 68 |
|---|---|---|
| | Range Sources | 64 |
| 6.7. | Appendix 7: List of Planned Laboratory Analytes with Reference | |
| | Increased Lipids from the Dyslipidemia SMQ (SMQ20000026) | 63 |
| 6.6. | Appendix 6: List of MedDRA Preferred Terms for Elevated or | |
| | Opportunistic Infections (POI) | 48 |
| 6.5. | Appendix 5: List of MedDRA Preferred Terms for Potential | |
| 6.4. | Appendix 4: Daily Diary Calculations | 45 |
| 6.3. | Appendix 3: Clinical Trial Registry Analyses | 45 |
| 6.2. | Appendix 2: Treatment Compliance | 44 |

# Version history

This Statistical Analysis Plan (SAP) for study J1P-MC-KFAH (KFAH) is based on the protocol dated 18Nov2020 and approved prior to unblinding.

Table KFAH.1. SAP Version History Summary

| SAP<br>Version | Approval<br>Date | Change | Rationale |
|----------------|------------------|----------------|------------------|
| 1 | | Not Applicable | Original version |

## 1. Introduction

Study J1P-MC-KFAH is an adaptive Phase 2, randomized, double-blind, placebo-controlled trial of LY3471851 (NKTR-358) in patients with moderately to severely active ulcerative colitis.

There are no changes to the analyses described in the protocol.

# 1.1. Objectives, Endpoints, and Estimands

| Objectives | Endpoints |
|---|---|
| Primary | |
| To determine whether LY3471851 is<br>superior to placebo in inducing clinical<br>remission at Week 12 in patients with<br>moderately to severely active ulcerative<br>colitis (UC) | The difference in the proportion of participants who achieve clinical remission based on MMS at Week 12 without permanently discontinuing treatment |
| Secondary | |
| To evaluate the efficacy of induction treatment with LY3471851 compared to placebo with respect to clinical, endoscopic, and histologic improvement | The difference between LY3471851 and placebo in the proportion of participants who have not permanently discontinued at Week 12 and have achieved at Week 12: clinical response endoscopic remission endoscopic response symptomatic remission symptomatic response histologic remission histologic-endoscopic mucosal healing |
| To evaluate the efficacy of maintenance | The difference between LY3471851 |
| treatment with LY3471851 compared to placebo with respect to clinical, | and placebo in the proportion of participants who were responders at |

| endoscopic, and histologic improvement | Week 12 (Week 12 Responders) and have not permanently discontinued at Week 52, who at Week 52 still have: clinical remission clinical response endoscopic remission endoscopic response symptomatic remission symptomatic response histologic remission histologic-endoscopic mucosal healing |
|---|---|
| To evaluate the efficacy of treatment with LY3471851 compared to placebo with respect to patient-reported outcomes and quality of life measures | <ul> <li>Comparison of mean changes from baseline to Week 12 and to Week 52 in scores for</li> <li>IBDQ</li> <li>Urgency NRS</li> <li>Abdominal Pain NRS</li> <li>Nocturnal Stools</li> <li>Bristol Stool Scale</li> <li>PGR-S</li> <li>Fatigue NRS</li> </ul> |
| To evaluate the PK of LY3471851 | Week 12 LY3471851 trough<br>concentrations |
| Tertiary/Exploratory | |
| CCI | |



Abbreviations: CC ; IBDQ = Inflammatory Bowel Disease Questionnaire; MMS = modified Mayo score, NRS = numeric rating scale; PGR-S = Patient's Global Rating of Severity; PK = pharmacokinetics; UC = ulcerative colitis; CC .

## **Primary estimand**

The primary clinical question of interest is: What is the intervention difference in successful response rate of clinical remission based on MMS at Week 12 of intervention in patients with moderately to severely active UC, where successful response is defined as patient who achieves clinical remission without discontinuing treatment, without increasing mandatory stable medications, and without taking prohibited medications prior to the time point of interest? The primary comparison will be assessed using a composite estimand strategy to address the intercurrent events.

The estimand is described by the following attributes:

Population: patients with moderately to severely active UC. Further details can be found in Section 3.

Endpoint: clinical remission based on MMS at Week 12 in MMS.

Treatment condition: the randomized treatment without rescue medication or change in background medication (treatment policy strategy). Further details on study interventions and concomitant, including rescue, interventions can be found in Section 6.

The 2 intercurrent events "intervention discontinuation for any reason" and "initiation of rescue intervention or change in background intervention" are both addressed by the treatment condition of interest attribute. There are no remaining intercurrent events.

Population-level summary: difference in proportion of participants achieving clinical remission at Week 12 between intervention conditions.

Rationale for estimand: The data collected after the treatment discontinuation or post-rescue medication will be categorized as nonresponder.

## **Secondary estimands**

1) Clinical response / endoscopic remission / endoscopic response / symptomatic remission / symptomatic response / histologic remission / histologic-endoscopic mucosal healing at Week 12

The secondary clinical question of interest is: What is the intervention difference in successful response rate of clinical response / endoscopic remission / endoscopic response / symptomatic remission / symptomatic response / histologic remission / histologic-endoscopic mucosal healing at Week 12 of intervention in patients with moderately to severely active UC, where successful response is defined as patient who achieves clinical response / endoscopic remission / endoscopic response / symptomatic remission / symptomatic response / histologic remission / histologic-endoscopic mucosal healing without discontinuing treatment, without increasing mandatory stable medications, and without taking prohibited medications prior to the time point of interest? The secondary comparisons will be assessed using a composite estimand strategy to address the intercurrent events.

The estimand is described by the following attributes:

Population: patients with moderately to severely active UC who have not permanently discontinued at Week 12 and have achieved at Week 12. Further details can be found in Section 3.

Endpoint: clinical response / endoscopic remission / endoscopic response / symptomatic remission / symptomatic response / histologic remission / histologic-endoscopic mucosal healing at Week 12.

Treatment condition: the randomized treatment without rescue medication or change in background medication (treatment policy strategy). Further details on study interventions and concomitant, including rescue, interventions can be found in Section 6.

The 2 intercurrent events "intervention discontinuation for any reason" and "initiation of rescue intervention or change in background intervention " are both addressed by the treatment condition of interest attribute. There are no remaining intercurrent events.

Population-level summary: difference in proportion of participants achieving clinical response / endoscopic remission / endoscopic response / symptomatic remission / symptomatic response / histologic remission / histologic-endoscopic mucosal healing at Week 12 between intervention conditions.

Rationale for estimand: The data collected after the treatment discontinuation or post-rescue medication will be categorized as nonresponder.

2) Clinical remission / clinical response / endoscopic remission / endoscopic response / symptomatic response / histologic remission / histologic-endoscopic mucosal healing at Week 52

The secondary clinical question of interest is: What is the intervention difference in successful response rate of clinical response / endoscopic remission / endoscopic response / symptomatic remission / symptomatic response / histologic remission / histologic-endoscopic mucosal healing at Week 52 of intervention in patients with moderately to severely active UC, where successful response is defined as patient who achieves clinical response / endoscopic remission / endoscopic response / symptomatic remission / symptomatic response / histologic remission / histologic-endoscopic mucosal healing without discontinuing treatment, without increasing mandatory stable medications, and without taking prohibited medications prior to the time point of interest?

The estimand is described by the following attributes:

Population: patients with moderately to severely active UC who were responders at Week 12, have not permanently discontinued at Week 52, have achieved at Week 52. Further details can be found in Section 3.

Endpoint: clinical remission / clinical response / endoscopic remission / endoscopic response / symptomatic response / histologic remission / histologic-endoscopic mucosal healing at Week 52.

Treatment condition: the randomized treatment without rescue medication or change in background medication (treatment policy strategy). Further details on study interventions and concomitant, including rescue, interventions can be found in Section 6.

The 2 intercurrent events "intervention discontinuation for any reason" and "initiation of rescue intervention or change in background intervention " are both addressed by the treatment condition of interest attribute. There are no remaining intercurrent events.

Population-level summary: difference in percentage of participants achieving clinical remission / clinical response / endoscopic remission / endoscopic response / symptomatic remission / symptomatic response / histologic remission / histologic-endoscopic mucosal healing at Week 52 between intervention conditions.

Rationale for estimand: The data collected after the treatment discontinuation or post-rescue medication will be categorized as nonresponder.

3) IBDQ / Urgency NRS / Abdominal Pain NRS / Nocturnal Stools / Bristol Stool Scale / PGR-S / Fatigue NRS

The secondary clinical question of interest is: What is the intervention difference in IBDQ / Urgency NRS / Abdominal Pain NRS / Nocturnal Stools / Bristol Stool Scale / PGR-S / Fatigue NRS at Week 12 and Week 52 of intervention in patients with moderately to severely active UC regardless of intervention discontinuation for any reason and regardless of initiation of rescue intervention or change in background intervention?

The estimand is described by the following attributes:

Population: patients with moderately to severely active UC. Further details can be found in Section 3.

Endpoint: IBDQ / Urgency NRS / Abdominal Pain NRS / Nocturnal Stools / Bristol Stool Scale / PGR-S / Fatigue NRS at Week 12 and Week 52.

Treatment condition: the randomized treatment without rescue medication or change in background medication (treatment policy strategy). Further details on study interventions and concomitant, including rescue, interventions can be found in Section 6.

The 2 intercurrent events "intervention discontinuation for any reason" and "initiation of rescue intervention or change in background intervention " are both addressed by the treatment condition of interest attribute. There are no remaining intercurrent events.

Population-level summary: difference in mean change in IBDQ / Urgency NRS / Abdominal Pain NRS / Nocturnal Stools / Bristol Stool Scale / PGR-S / Fatigue NRS at Week 12 and Week 52 between intervention conditions.

Rationale for estimand: The data collected after the treatment discontinuation or post-rescue medication will not represent the true efficacy effects.

## 1.2. Study Design

Study KFAH is an adaptive Phase 2 multicenter, randomized, double-blind, placebo-controlled, parallel-group study to evaluate the efficacy and safety of multiple dose levels of LY3471851 in adult patients with moderately to severely active UC. Enrolled study participants will have either

- an inadequate response to, loss of response to, or be intolerant to corticosteroid or immunomodulator therapy for UC (termed "conventional-failed"), or
- an inadequate response to, loss of response to, or are intolerant to biologic or JAK inhibitor therapy for UC (termed "advanced therapy-failed").

## **Study Stages**

This adaptive study has two stages.

Stage 1: Approximately 100 participants will be randomly assigned to one of three treatment groups, including placebo. Interim analyses will be conducted for safety, dosing tolerability, and efficacy. These interim analyses will determine the doses to be used in Stage 2.

**Note:** Participants enrolled during Stage 1 of the study will remain on their randomly assigned Stage 1 doses. Their doses will be changed only if necessary due to safety reasons or due to their clinical response status at the end of Stage 1.

Stage 2: Approximately 100 additional study participants will be enrolled and randomly assigned to study treatment groups as well as placebo. The treatment doses used in Stage 2 may include any of the doses used in Stage1, as well as one or more additional LY3471851 doses, not exceeding1800 µg. The Stage 2 LY3471851 treatment doses will be determined by the sponsor based on results of the Stage 1 interim analyses and recommendations of the sponsor's IAC. A small group of sponsor personnel having pre-identified roles and no contact with investigative sites may review the IAC recommendation and may also review unblinded data in order to further assess the recommendation. The IAC charter that describes the process for internal decision-making and action plan will be provided.

Thus, whereas Stage 1 will have three treatment groups (including placebo), Stage 2 could have more treatment groups or fewer (including placebo).

The sponsor intends for the transition from Stage 1 to Stage 2 to be seamless, with participant screening and enrollment activities occurring continuously in the transition period. The study IWRS will allocate newly enrolling participants to groups according to the Stage 1 randomization ratio until the Stage 2 groups have been decided upon and implemented. The randomization ratios are described in Section 1.2.1.

### **Study Periods**

This study has multiple periods.

Screening period

This period begins with Visit 1, which occurs 5 weeks (or less) before the planned randomization visit. A participant's screening evaluations must be completed and reviewed to confirm the participant's eligibility before randomization and dosing occurs at Visit 2.

## Blinded induction and blinded maintenance periods

The double-blind, placebo-controlled, 12-week induction treatment period begins at Visit 2. Dosing, sample collection, and assessments continue Q2W, as shown in the SOA in the protocol. Between Week 12 and Week 14, based on samples and assessments collected at Week 12, participants will be classified as either "Week 12 Responders" or "Week 12 Nonresponders" based on the "clinical response" criteria defined in the protocol.

- "Week 12 Responders" will continue to receive their same randomly assigned treatment throughout the blinded 40-week Maintenance Period, with the final dose occurring at Week 50 and the last maintenance assessments and sample collections at Week 52.
- "Week 12 Nonresponders" will enter the Extension Induction and Extension Maintenance Periods.

## Extension induction and maintenance periods

Beginning at Week 14, participants who were classified as Week 12 Nonresponders will receive the high dose (DD µg) of LY3471851 Q2W, unless a lower dose is selected for Stage 2 based on interim analyses.

Between Week 26 and Week 28, based on samples and assessments collected at Week 26, these participants will again be classified according to their clinical response status based on MMS (responder or nonresponder).

- Participants who are classified as responders based on the samples and assessments at Week 26 will continue to receive LY3471851 Q2W as maintenance through the remainder of the study. These participants have their final dose at Week 50 and their last maintenance assessments and sample collections at Week 52.
- Participants who are classified as nonresponders based on the Week 26 samples and assessments will be permanently discontinued from study drug when his/her status as a nonresponder has been determined; such participants will enter the post-treatment follow-up period.

#### Post-treatment follow-up period

All participants will have a post-treatment follow-up visit (Visit 801) for safety assessments. Visit 801 occurs approximately 6 weeks after the Week 52 visit. The last dose of study drug is given at Week 50. Thus, participants will have been withdrawn from study drug for approximately 8 weeks at Visit 801. Participants who were positive for anti-HBc at screening will have one additional post-treatment follow-up visit (Visit 802).

#### Early discontinuation

Participants who permanently discontinue the study drug early or withdraw from the study will undergo early termination procedures, including an ETV and the post-treatment follow-up visits specified in the SoA.

Figure KFAH.1 and Figure KFAH.2 show the study design.



Abbreviations: D = day; DNA = deoxyribonucleic acid; ETV = early termination visit; HBV = hepatitis B virus; LY= LY3471851; Q2W = every 2 weeks; W = Week; w = weeks.

Figure KFAH.1. Study Schematic (Induction and Maintenance Periods)



Abbreviations: DNA = deoxyribonucleic acid; ETV = early termination visit; HBV = hepatitis B virus; Q2W = every 2 weeks; W = Week; w = weeks.

Note: The extension dose could be lower than CCI µg LY3471851, based on interim analyses.

Figure KFAH.2. Study Schematic (Nonresponder Extension Periods)

## 1.2.1. Method of Assignment to Treatment

Patients who meet all criteria for enrollment will be randomized to treatment at the baseline visit. Assignment to treatment groups will be determined by a computer-generated random sequence using an interactive web-response system (IWRS), and then the site will be responsible for administering the treatment to the patients.

During Induction Period in Stage 1, approximately 100 participants will be randomized to 1 of 3 treatment groups in a 2:2:1 ratio:

- CC μg LY3471851 Q2W SC,
- μg LY3471851 Q2W SC, or
- placebo.

During Induction Period in Stage 2, up to approximately 100 additional participants will be randomized. The number of treatment groups and randomization ratio for Stage 2 will be determined and documented based on the last interim analysis of Stage 1. This decision making will occur following Stage 1, and the choice in allocation ratio including placebo may be adjusted to achieve the planned allocation across treatment arms.

The randomization will be stratified based on the following factors:

- previous advanced therapy failure status (yes/no)
- baseline corticosteroid use (yes/no), and
- baseline disease activity (MMS: [4 to 6] or [7 to 9]).

After the Induction Period, participants enter either Maintenance Period or Extension Induction and Extension Maintenance Periods, based on samples and assessments collected at Week 12, as described in Section 1.2.

## 2. Statistical Hypotheses

The primary objective is to demonstrate that LY3471851 is superior to placebo in achieving clinical remission at Week 12. Thus, the null hypothesis to be tested in relation to the primary estimand is that LY3471851 is not different from placebo with respect to the achievement of clinical remission at Week 12.

## 2.1. Multiplicity Adjustment

Multiplicity adjustment will not be employed in the analysis for this study.

## 3. Analysis Sets

Table KFAH.2 describes the populations planned for use in the analyses. The mITT population, as defined below, will be used in analyses of efficacy and PRO, unless otherwise noted in the SAP.

Table KFAH.2. Analysis Populations

| Population | Description |
|---|---|
| ITT Population | All randomized participants. Participants will be analyzed according to the treatment to which they were assigned. |
| mITT Population | All randomized participants who receive at least 1 dose of study treatment (regardless of whether the participant fails to receive the correct treatment, or otherwise fails to follow the protocol). Participants will be analyzed according to the treatment to which they were assigned. |
| Safety Population | Same as mITT population |
| Pharmacokinetic Evaluable | All participants who receive at least 1 dose of investigational product and have sufficient blood sampling to allow for pharmacokinetic evaluation. |

Abbreviations: GCP = Good Clinical Practice; ITT = intent-to-treat; mITT = modified intent-to-treat; SAP = statistical analysis plan.

Analyses of the maintenance dosing period and the extension periods will be based on the corresponding enrolled population as described in the table above.

## 4. Statistical Analyses

### 4.1. General Considerations

This SAP is intended to describe the analyses of all objectives, as well as safety assessments, for study KFAH.

Statistical analysis of this study will be the responsibility of Eli Lilly and Company (hereafter Lilly) or its designee. For primary and key secondary objectives, statistical analyses will be performed using SAS® Enterprise 7.1 or higher, SAS® Version 9.4 or higher, or RStudio Server Pro Version R.3.6.3. or higher.

Efficacy analyses will be conducted on the mITT population. Safety analyses will be conducted on the Safety population (same as mITT population, as described in Section 3). The efficacy analysis of the primary endpoint and secondary endpoints will be repeated for ITT population. Additional safety analyses may be performed as deemed appropriate.

The baseline modified Mayo Score (MMS) is calculated from valid daily diary entries obtained prior to endoscopy during the screening period and the endoscopic appearance of the mucosa at this screening endoscopy. For other efficacy, health outcome and safety assessments, baseline is defined as the last non-missing assessment recorded on or prior to the date of the randomization visit (Visit 2).

Any change to the data analysis methods described in the protocol will require an amendment ONLY if it changes a principal feature of the protocol. Any other change to the data analysis methods described in the protocol and the justification for making the change will be described in the clinical study report. Additional exploratory analyses of the data will be conducted as deemed appropriate.

Not all displays and analyses described in this SAP will necessarily be included in the CSR. Not all displays will necessarily be created as a "static" display. Some displays may be incorporated as interactive display tools instead of or in addition to a static display. Any display described in this SAP and not provided in CSR would be available upon request.

### 4.1.1. Analysis Methods

Continuous data will be summarized in terms of the number of observations, mean, standard deviation (SD), median, minimum, and maximum. The minimum and maximum will be reported to the same number of decimal places as the raw data recorded in the database. The mean and median will be reported to one more decimal place than the raw data recorded in the database. The SD will be reported to two more decimal places than the raw data recorded in the database. In general, the maximum number of decimal places reported shall be four for any summary statistic.

Categorical data will be summarized in terms of the number of patients providing data at the relevant time point (n), frequency counts and percentages. Percentages will be presented to one decimal place. Percentages will be calculated using n (the number of observations with non-missing values) as the denominator.

Unless otherwise specified, analysis of hypotheses will be tested without multiplicity control at a significance level of 0.05. A 2-sided 95% CI will be provided along with the p-value. P-values

which are greater than or equal to 0.001, and less than or equal to 0.999, will be presented to three decimal places. All other p-values which are less than 0.001 will be presented as '<0.001', while p-values greater than 0.999 will be presented as '>0.999'. CIs will be presented to one more decimal place than the raw data.

Unless otherwise specified, variables will be analyzed in the original scale on which they are measured. However, if it is deemed more statistically appropriate, a transformation, such as to the logarithmic scale, may be applied before analysis. The parametric approach will be employed by default for statistical analysis except when nonparametric analysis, such as by a rank-based method, is considered to be more fitting.

For assessments of the primary endpoint, other categorical (binary) efficacy, the Cochran-Mantel-Haenszel (CMH) chi-square test will be used to compare the treatment groups with the following factors:

- previous advanced therapy failure status (yes/no)
- baseline corticosteroid use (yes/no)
- baseline disease activity (MMS: [4 to 6] or [7 to 9]), and
- region (North America/Europe/Other).

The CMH chi-square p-value and the relative risk along with its 2-sided CI will be provided. In addition, the absolute treatment difference in proportions will be provided along with the 2-sided CI estimate. The differences between each treatment group and placebo will also be tested separately using a logistic regression model that controls for at least previous advanced therapy failure status (yes/no) and corticosteroid use (yes/no). If deemed necessary, additional analyses of categorical efficacy variables may be conducted to address sparse data and/or small sample sizes.

Treatment comparisons of continuous efficacy and health outcome variables with multiple postbaseline time points will be made using MMRM analysis. The MMRM will include the following effects and covariates:

- treatment group
- previous advanced therapy failure status (yes/no)
- corticosteroid use (yes/no)
- disease activity (MMS: [4 to 6] or [7 to 9]) at baseline)
- region (North America/Europe/Other)
- baseline value in the model
- visit, and
- the interactions of treatment-by-visit and baseline-by-visit as fixed factors.

The covariance structure to model the within-participant errors will be unstructured. If the unstructured covariance matrix results in a lack of convergence, the heterogeneous Toeplitz covariance structure, followed by the heterogeneous autoregressive covariance structure, will be used. The first structure to yield convergence will be used for inference. The Newton-Raphson with ridging optimization technique will be used to aid with convergence. The Kenward-Roger

method will be used to estimate the denominator degrees of freedom. Type III sums of squares for the LS means will be used for the statistical comparison; the 95% CI will also be reported. Treatment group comparisons with placebo at Week 12 and all other appropriate time points will be tested.

Treatment comparisons of continuous efficacy and health outcome variables with a single postbaseline time point will be made using ANCOVA with the following in the model:

- treatment group
- previous advanced therapy failure status (yes/no)
- corticosteroid use (yes/no)
- disease activity (MMS: [4 to 6] or [7 to 9]) at baseline)
- region (North America/Europe/Other), and
- baseline value.

Type III sums of squares for LS means will be used for statistical comparison between treatment groups. The LS mean difference, standard error, p-value, and 95% CI, unless otherwise specified, will also be reported.

## 4.1.2. Handling of Dropouts or Missing Data

Intercurrent events (FDA 2017) are events which occur after the study intervention initiation and make it impossible to measure a variable or influence how it should be interpreted. Examples of such events include treatment discontinuation due to death or adverse events (AEs), rescue treatment, and loss to follow-up. The missing data handling methods described below describe how intercurrent events will be used for the different estimands.

### 4.1.2.1. Non-Responder Imputation (NRI)

The primary outcome is the proportion of patients with clinical remission at Week 12. For this and other categorical efficacy endpoints (for example, clinical remission (week 52), clinical response (week 12, 52), and endoscopic remission (week 12, 52)), non-responder imputation (NRI) will be used for missing clinical assessment values. Specifically, all patients who discontinue from the study at any time prior to week 12 for any reason or fail to have an adequate week 12 efficacy assessment will be considered a non-responder at week 12. Patients who discontinue from the study for any reason at any time prior to week 52 after having enrolled into the Maintenance Period or fail to have an adequate week 52 efficacy assessment, will be considered a non-responder at week 52.

The NRI may be applied at any time point specified for analysis.

## 4.1.2.2. Mixed-Effects Model for Repeated Measures

For the continuous secondary and exploratory efficacy and health outcome variables, MMRM analyses will be the main method to mitigate the impact of missing data. This approach assumes that missing observations are missing-at-random (missingness is related to observed data) during the study and takes into account both the missingness of data and the correlation of the repeated measurements.

All continuous endpoints will utilize MMRM to patients who permanently discontinued study drug or who were rescued.

### 4.1.2.3. Modified Baseline Observations Carried Forward (mBOCF)

For patients discontinuing investigational product due to an AE, the baseline observation for the endpoint will be carried forward to the corresponding visit for all missing observations after the patient discontinued study treatment. For patients discontinuing investigational product for any other reason, the last non-missing postbaseline observation before discontinuation will be carried forward to the corresponding visit for all missing observations after the patient discontinued. For all patients with sporadically missing observations prior to discontinuation, the last non-missing observation before the sporadically missing observation will be carried forward to the corresponding visit. Randomized patients without at least 1 postbaseline observation will not be included for evaluation with the exception of patients discontinuing study treatment due to an AE.

The mBOCF method is based on an estimand that handles the intercurrent event of discontinuing study drug due to an AE by defining the patient as not receiving any benefit from study drug after the event. That is the patient is defined as reverting back to baseline regardless of any continuing efficacy benefits they may still have received after the event. For other intercurrent events (e.g., rescue treatment and discontinuation due to reasons other than an AE) or sporadic missingness the "while on treatment" strategy is applied. That is, the endpoint is defined as the last observed value at or before the visit of interest before the patient discontinued study treatment.

## 4.2. Participant Dispositions

A detailed description of participant disposition will be provided, including a summary of the number and percentage of participants entered into the study and randomized, the number and percentage of participants who complete the study or discontinue, both overall and by reason for discontinuation, and the frequency and percentage of patients who discontinue study treatment. A summary of important protocol deviations will be provided.

# 4.3. Primary Endpoint Analysis

### 4.3.1. Definition of endpoint

Rate of clinical remission at Week 12 is the primary efficacy outcome for this study and will be analyzed using the mITT population.

Clinical remission is defined as achieving a rectal bleeding (RB) subscore of 0, and stool frequency subscore (SF) of 0, or 1 with a decrease of  $\geq$ 1 point from baseline, and endoscopic (ES) subscore of 0 or 1, excluding friability. SF and RB subscores are calculated by averaging and rounding the 4-point daily scores over 3 days as described in 6.6.

### 4.3.2. Main analytical approach

The primary objective of this study is to test the hypothesis that treatment with LY3471851 is superior to placebo in inducing clinical remission at Week 12 in patients with moderate to severe ulcerative colitis (UC).

The rates of clinical remission and non-remission will be summarized by treatment group and by the stratification factors, previous advanced therapy failure status (yes/no), baseline corticosteroid use (yes/no), baseline disease activity (MMS: [4 to 6] or [7 to 9]), and region (North America/Europe/Other).

The primary analysis will use the CMH chi-square test to compare LY3471851 to placebo at Week 12. The stratification factors used for CMH test are (a) previous advanced therapy failure status (yes/no), (b) baseline corticosteroid use (yes/no), (c) baseline disease activity (MMS: [4 to 6] or [7 to 9]), and (d) region (North America/Europe/Other). See Section 4.1.1 for details on the methods to be used to test the differences between each active treatment arm and placebo.

Ninety five percent confidence interval along with the p-value for the difference in proportions (LY arm – placebo) for each pairwise comparison will be obtained. For a pairwise comparison, if p-value is less than 0.05, then that LY arm will be considered to be superior to placebo.

A composite strategy is proposed for other intercurrent events including discontinuing study intervention, taking prohibited medications or increase the dose of mandatory stable medications. The NRI methodology described in Section 4.1.2.1 will be applied when any of these events occur.

## 4.3.3. Bayesian Model Averaging

A Bayesian model averaging will be performed for additional analysis of the clinical remission at Week 12. A Bayesian model averaging (BMA) approach will be used to estimate the dose response relationship. This Bayesian model averaging approach is the Bayesian analog of the MCP-MOD methodology (Bretz et al., 2005), and "the Qualification of the MCP-Mod procedure" (FDA, 2015) is supportive in the use of MCP-MOD or Bayesian model averaging to assist in dose selection decisions.

Bayesian model averaging is a general mixture distribution, where each mixture component is a different parametric model. Prior weights are placed on each model and the posterior model weights are updated based on how well each model fits the data. Let  $\mu(d)$  represent the mean of the dose response curve at dose d,  $y = \{y_1, ..., y_n\}$  be the observed data, and  $m \in \{1, ..., M\}$  be an index on the M parametric models described below. Then the posterior of the dose response curve,  $\mu(d)$ , of the Bayesian model averaging model is

$$p(\mu(d) \mid y) = \sum_{m=1}^{M} p(\mu(d) \mid y, m) p(m \mid y)$$
$$p(m \mid y) = \frac{p(y \mid m) p(m)}{\sum_{m^*} p(y \mid m^*) p(m^*)}$$

where  $p(\mu(d) \mid y, m)$  is the posterior mean dose response curve from model m,  $p(m \mid y)$  is the posterior weight of model m,  $p(y \mid m)$  is the marginal likelihood of the data under model m, and p(m) is the prior weight assigned to model m. In cases where  $p(y \mid m)$  is difficult to compute, Gould (2019) propose using the observed data's fit to the posterior predictive distribution as a surrogate in calculating the posterior weights; this is the approach used in this analysis.

## 4.3.3.1. BMA Analysis and Reporting

BMA will be executed for the proportion of participants who achieve clinical remission at Week 12.

BMA analysis will be summarized by dose and provide

- Observed response
- BMA estimated
  - Mean response
  - o Standard error and standard deviation of the mean response
  - o 2.5% and 97.5% quantiles
  - Summaries of posterior probability of LY PBO treatment effect, i.e.,
     Pr(LY PBO > EOI) where EOI is effect of interest
- Plot that includes observed response, BMA estimated response, 2.5% and 97.5% posterior quantiles

BMA analysis will be summarized by component and model parameter and provide

- Posterior mean
- Standard error and standard deviation of the posterior mean
- 2.5% and 97.5% posterior quantiles of the posterior distribution
- Convergence diagnostics
- Effective sample size
- Prior distributions
- Plot of the fitted BMA
- Plot of the BMA components

## 4.4. Secondary Endpoints Analyses

## 4.4.1. Secondary Efficacy Endpoints

### 4.4.1.1. Definition of Endpoints

In the analyses of secondary efficacy outcomes, no adjustments for multiple testing will be performed unless otherwise specified.

The efficacy assessments of secondary endpoints are shown in the following table:

Table KFAH.3. Efficacy Assessments

| Clinical Remission | SF subscore = $0$ , or SF = $1$ , and RB subscore = $0$ , and ES = $0$ or $1$ , excluding friability. |
|---|---|
| Clinical Response | A decrease in the MMS of $\geq 2$ points and $\geq 30\%$ decrease from baseline, and a decrease of $\geq 1$ point in the RB subscore from baseline or a RB score 0 or 1. |
| Endoscopic Remission | Mayo ES = 0 or 1, excluding friability. |

| Endoscopic Response | A decrease in the Mayo ES of ≥1 point compared to baseline. |
|---|---|
| Symptomatic Remission | $SF = 0$ , or $SF = 1$ with a decrease of $\geq 1$ point from baseline, and $RB = 0$ . |
| Symptomatic Response | ≥30% decrease from baseline in the composite clinical endpoint of the sum of SF and RB subscores. |
| Histologic Remission | Geboes score <2 or Geboes subscores = 0 for Grade 2a, 2b, 3, 4, and 5. |
| Histologic-Endoscopic<br>Mucosal Healing | Geboes scroe <2 and endoscopic remission. |

Abbreviations: ES = endoscopic subscore; MMS = modified Mayo score; RB = rectal bleeding; SF = stool frequency.

## 4.4.1.2. Secondary Efficacy Endpoints for the Induction Period

Secondary efficacy endpoints for the induction dosing period for participants who have not permanently discontinued at Week 12 and have achieved at Week 12 include clinical response, endoscopic remission, endoscopic response, symptomatic remission, symptomatic response, histologic remission, and histologic-endoscopic mucosal healing at Week 12.

Analyses will be performed as per the methodology described in Section 4.1.1.

The mITT population will be used for the secondary efficacy outcome analyses.

### 4.4.1.3. Secondary Efficacy Endpoints for the Maintenance Period

Secondary efficacy endpoints for the maintenance period for participants who were responder per IWRS at Week 12, have not permanently discontinued at Week 52, and have achieved at Week 52 include clinical remission, clinical response, endoscopic remission, endoscopic response, symptomatic remission, symptomatic response, histologic remission, and histologic-endoscopic mucosal healing at Week 52.

Analyses will be performed as per the methodology described in Section 4.1.1.

The mITT population will be used for the secondary efficacy outcome analyses.

### 4.4.2. Secondary Health Outcome Endpoints

The following are patient-reported outcome instruments collected using a participant eDiary:

- Rectal Bleeding
- Stool Frequency
- Nocturnal Stool
- Bristol Stool Scale

- Urgency NRS
- Abdominal Pain NRS
- Fatigue NRS, and
- PGR-S

The following are patient-reported outcome instruments collected electronically:

- PGI-C and
- IBDQ

Where appropriate, the total scores and sub-totals for individual dimensions collected will be summarized with means and 95% CIs by time point and by treatment group. The summary table will also include the change from baseline scores wherever applicable. The mean raw scores and mean change from baseline scores with corresponding 95% CIs will be presented graphically by treatment group and in a longitudinal fashion.

The ITT population will be used for all health outcome analyses

Mean change from baseline will be summarized by treatment group.

## 4.4.3. Bioanalytical and Pharmacokinetic/Pharmacodynamic Methods

PK/PD analyses to address secondary and exploratory objectives of this study will be described by Lilly in separate PK/PD analysis plans. Conduct of the PK/PD analyses will be the responsibility of Eli Lilly and Company.

The PK/PD analyses will be initiated up to approximately three weeks before the planned database lock dates. All analyses will be performed by unblinded Lilly PK personnel, who are unblinded to subject treatment assignments to support dose adjustments. Results from the PK/PD analyses will not be shared with site or blinded study team personnel prior to the respective database lock.

## 4.5. Tertiary/Exploratory Endpoints Analyses





## 4.6. Safety Analyses

All safety data will be descriptively summarized by treatment groups and analyzed based on the safety population as defined in Section 3. The safety analyses include AEs, safety in special groups and circumstances, including Adverse Events of Special Interest (AESI), laboratory analytes, QIDS-SR16, C-SSRS, ECGs, and vital signs. The duration of exposure will also be summarized. The categorical safety measures will be summarized using incidence rates and analyzed by Fisher's exact test. The mean change in the continuous safety measures including vital signs, QIDS-SR16, physical characteristics, and laboratory values will be summarized by visits and analyzed by ANCOVA, with treatment and baseline values in the model. More details are provided in subsequent sections.

For specific events of special interest (see Section 4.6.3 for more details), an incidence rate, IR per 100 patient-years of observation (PYO), will be provided. Patient-years of observation will be calculated as the sum of all patient observation time in the treatment group. For a patient with an event, the observation time will be censored at the event date; for a patient without the event, the observation time will be counted until the patient's last treatment dose date plus 30 days or the patient's last visit, whichever occurs first. Only events that occur within 30 days after the patient's treatment discontinuation date will be considered.

See formula as follows:

$$PYO = \sum_{pt \ w \ event} \frac{event \ start \ date - first \ trt \ dose \ date + 1}{365.25} + \sum_{pt \ w/o \ event} \frac{last \ observation \ date - first \ trt \ dose \ date + 1}{365.25}$$

Incidence rate will be calculated as follows:

$$IR = \frac{unique\ number\ of\ patients\ with\ event}{PYO} \times 100$$

For each IR provided, a 95% CI will be calculated based on the Poisson distribution. Treatment group comparisons based on IR will be provided based on the incidence rate difference (IRD) together with its 95% CI.

Not all displays described in this section will necessarily be included in the CSRs. Any display described and not provided in the CSR would be available upon request. Not all displays will necessarily be created as a "static" display. Some may be incorporated into interactive display tools instead of or in addition to a static display. Any display created interactively will be included in the CSR if deemed relevant to the discussion.

#### 4.6.1. Extent of Exposure

Duration of exposure to study treatment (defined as time since first injection of study treatment in days) will be summarized by treatment group during the Induction Period, the Maintenance Period, and the Extension Period.

Duration of exposure during the Induction Period for the Safety Population will be calculated as:

(Disposition date (for those who have discontinued the Induction Period), OR Maintenance/Extension Start date -1 (for those who have completed the Induction Period), OR Date of last study visit in the Induction Period (for those who are still being treated in the Induction Period) – Date of first injection of study treatment + 1)

Duration of exposure during the Maintenance Period will be calculated as:

(Disposition date (for those who have discontinued the Maintenance Period), OR Date of last study visit in the Maintenance Period (for those who are still being treated in the Maintenance Period) – Date of the Visit 10 injection of study treatment + 1)

Duration of exposure to LY3471851 during the Extension Period will be calculated as:

(Disposition date (for those who have discontinued the Extension Period), OR Date of last study visit in the Extension Period (for those who are still being treated in the Extension Period) — Date of the Visit 10 injection of study treatment + 1)

Duration of exposure to LY3471851 for the combined Induction Period and Maintenance Period will be calculated as:

(Disposition date (for those who have discontinued the Maintenance Period), OR Date of last study visit in the Maintenance Period (for those who are still being treated in the Maintenance Period)—Date of first injection of LY3471851 + 1)

Duration of exposure to LY3471851 for the combined Induction Period and Extension Period will be calculated as:

(Disposition date (for those who have discontinued the Extension Period), OR Date of last study visit in the Extension Period (for those who are still being treated in the Extension Period)—Date of first injection of LY3471851 + 1)

The date of first injection of LY3471851 is defined in Table KFAH.4

| | Visit of first LY3471851 |
|---|---|
| All patients randomized to LY3471851 (regardless of Week 12 response status) | Week 0 (Visit 2) |
| Week 12 Inadequate Responders originally randomized to placebo and assigned to LY3471851 at Visit 10 | Week 14 (Visit 10) |

Table KFAH.4. First Injection of LY3471851 by Treatment Group

Descriptive statistics (n, mean, SD, minimum, first quartile, median, third quartile, and maximum) will be provided for patient-days of exposure and the frequency of patients falling into different exposure ranges will be summarized. Exposure ranges are as follows:

- $>0, \ge 4$  weeks,  $\ge 12$  weeks, and  $\ge 52$  weeks.
- >0 to <4 weeks, >4 weeks to <12 weeks, >12 weeks to <52 weeks, and >52 weeks.

Additional exposure ranges may be considered if necessary.

A by-patient listing of exposure duration will be provided.

Patients who had dose modification will be grouped under the randomized treatment arm and will not be grouped by the modified dose amount.

No inferential analysis for comparison between treatment arms will be performed.

#### 4.6.2. Adverse Events

#### 4.6.2.1. Adverse Events

Adverse events are recorded in the eCRF. Each AE will be coded to SOC and PT, using the *Medical Dictionary for Regulatory Activities* (MedDRA) version that is current at the time of database lock. Severity of AEs is recorded as mild, moderate, or severe.

Treatment-emergent adverse events (TEAEs) are defined as events that either first occurred or worsened in severity after the first dose of study drug and the earliest of the visit study drug disposition date or the last visit date during the treatment period, whichever occurred first, and up to 30 days after study treatment discontinuation. The MedDRA Lowest Level Term (LLT) will be used in defining which events are treatment-emergent. The maximum severity for each LLT during the baseline period until the first dose of the study medication will be used as baseline. If an event is preexisting during the baseline period, but it has missing severity, and the event persists during the treatment period or up to 30 days after treatment discontinuation, then the baseline severity will be considered mild for determining any postbaseline treatment-emergence (i.e., the event is treatment-emergent unless the severity is coded mild at postbaseline). If an event occurring postbaseline has a missing severity rating, then the event is considered treatment-emergent. Should there be insufficient data for an AE start date to make this comparison (e.g., the AE start year is the same as the treatment start year, but the AE start month and day are missing), the AE will be considered treatment-emergent. For events occurring on the day of the first dose of study treatment, the day of the onset of the event will

both be used to distinguish between pretreatment and posttreatment in order to derive treatmentemergence.

In general, summaries will include the number of patients in the safety population (N), frequency of patients experiencing the event (n), and relative frequency (i.e., percentage; n/N\*100).

In an AE overview table, the number and percentage of patients in the safety analysis set who experienced death, a serious adverse event (SAE), any TEAE, permanent discontinuation from study drug due to an AE, or a severe TEAE will be summarized by treatment group.

The number and percentage of patients with TEAEs will be summarized by treatment group in 2 formats listed below. For events that are gender specific, the denominator and computation of the percentage will only include patients from the given gender.

- by MedDRA PT nested within SOC with SOCs ordered alphabetically, and events ordered within each SOC by decreasing frequency in the LY3471851 1800µg treatment group.
- by MedDRA PT with events ordered by decreasing frequency in the LY3471851 1800μg treatment group.

Adverse events leading to permanent discontinuation of study drug and AEs leading to temporary interruption of study drug will also be summarized by treatment group using MedDRA PT nested within SOC. Events will be ordered by decreasing frequency within SOC in the LY3471851 1800µg treatment group.

A summary of temporary interruptions of study drug will also be provided, showing the number of patients who experienced at least 1 temporary interruption and the number of temporary interruptions per patient with an interruption. Further, the duration of each temporary interruption (in days) and the cumulative duration of dose interruption (in days) using basic descriptive statistics (n, mean, SD, minimum, first quartile, median, third quartile, and maximum) will be displayed.

Common TEAEs are defined as TEAEs that occurred in ≥1% (before rounding) of patients in any treatment group including placebo. The number and percentage of patients with common TEAEs will be summarized by treatment using MedDRA PT ordered by decreasing frequency in the LY3471851 1800µg treatment group.

The number and percentage of patients with TEAEs will be summarized by maximum severity by treatment using MedDRA PT ordered by decreasing frequency for the common TEAEs. For each patient and TEAE, the maximum severity for the MedDRA level being displayed is the maximum postbaseline severity observed from all associated LLTs mapping to that MedDRA PT.

#### 4.6.2.2. Serious Adverse Events

An individual listing of all AEs including preexisting conditions will be provided. A separate listing will include AEs that led to permanent discontinuation from the study drug. In addition, a listing of AEs that occur more than 30 days after study treatment discontinuation will be provided.

With the International Conference on Harmonisation (ICH) E2A guideline, a SAE is any AE that results in 1 of the following outcomes:

- death
- initial or prolonged inpatient hospitalization
- a life-threating experience (that is, immediate risk of dying)
- persistent or significant disability/incapacity
- congenital anomaly/birth defect
- considered significant by the investigator for any other reason

The number and percentage of patients who experienced any ICH-defined SAE will be summarized by treatment group during the treatment and follow-up periods using MedDRA PT nested within SOC. Events will be ordered by decreasing frequency within SOC in the LY3471851 1800µg treatment group. In addition, the SAEs will be summarized by treatment group using MedDRA PT without SOC. An individual listing of all SAEs will be provided.

## **4.6.3.** Adverse Events of Special Interest

#### **4.6.3.1. Infections**

Infections will be defined using all PTs from the MedDRA Infections and Infestations SOC. Serious infection will be defined as all the infections that meet the SAE criteria.

The number and percentage of patients with TEAEs of infections, serious infections, and infections resulting in study drug discontinuation will be summarized by treatment group using MedDRA PTs.

The number and percentage of patients with TEAEs of infections by maximum severity will be summarized by treatment group using MedDRA PTs.

For infections of special interest (serious infections, potential opportunistic infections [POIs], herpes zoster, and herpes simplex), the IR (for detail, see Section 4.6) and 95% CI will be calculated.

Treatment-emergent infectious events will be reviewed in context of other clinical and laboratory parameters. A listing of patients experiencing treatment-emergent infectious AEs will be provided. The listing will include patient demographics, treatment group, treatment start and stop dates, infectious event, event start and stop dates, total leukocytes, total lymphocytes, absolute neutrophils, event seriousness, and event outcome.

The infectious TEAE will be further analyzed in terms of potential opportunistic infection, herpes zoster, and herpes simplex. A summary of hepatitis B virus (HBV) deoxyribonucleic acid (DNA) monitoring results and association between infection and neutropenia/lymphopenia will also be provided in the context of infections.

## **Potential Opportunistic Infections**

Potential opportunistic infections will be identified according to 2 different approaches.

First, POIs will be identified from TEAEs based on a Lilly-defined list of MedDRA PTs shown in 6.8. These PTs are a subset of terms from the Infections and Infestations SOC.

Second, a list of all the infection details captured from the infection-specific eCRF (including primary/secondary infecting organism and infection site) will be provided. Of note, the infecting organism that was entered as free text by the investigator (instead of as a selection from the pull-down list) will also be provided.

The summary analysis of POIs identified using the 2 approaches above will be provided. Each case meeting the case definition for an opportunistic infection will be summarized by PT nested under infection pathogen. Events will be ordered by decreasing frequency of pathogen nested under pathogen species (mycobacteria, bacteria, fungal, viral, parasites). The order of frequency will be determined using the LY3471851 1800µg group.

Potential opportunistic infections identified through these approaches will be combined in 1 list for medical assessment for final classification of whether the case definition was met according to the consensus paper after database lock (i.e., Winthrop 2015). An additional summary may be conducted based on medical assessment.

#### **Herpes Zoster**

A summary table of herpes zoster will be provided. Herpes zoster will be defined based on the MedDRA PTs as listed under Herpes zoster (any form) (II) in 6.8, excluding Varicella virus text (10070444). The summary table will also include event maximum severity, seriousness, whether resulting in temporary study drug interruption, whether resulting in study drug discontinuation, whether treated with antiviral medication, and event outcome.

If a patient has more than 1 event of herpes zoster, the event with the maximum severity will be used in these summary tables. If more than 1 event of herpes zoster occurs with the same severity, the event with the longest duration will be used in the summary table.

#### **Herpes Simplex**

A summary analysis of herpes simplex will be provided. Herpes simplex will be defined based on the MedDRA PTs as listed under Herpes simplex (invasive disease only) (IV) in 6.8. The summary table will include event maximum severity, seriousness, whether resulting in temporary study drug interruption, whether resulting in study drug discontinuation, and whether treated with antiviral medication. Antiviral medication will be selected based on ATC code level 2 "antiviral for systemic use."

If a patient has more than 1 event of herpes simplex, the event with the maximum severity will be used in these summary tables. If more than 1 event of herpes simplex occurs with the same severity, the event with the longest duration will be used in the summary table.

#### **HBV DNA**

A listing of patients with detectable HBV DNA will be provided.

HBV DNA status (not detectable, detectable but not quantifiable [ie, <29 IU/mL], quantifiable [ie, ≥29 IU/mL]) will be summarized by treatment group stratified by baseline HBV serology status, specifically:

- HBsAb-/HBcAb-
- HBsAb+/HBcAb-

- HBsAb+/HBcAb+
- HBsAb-/HBcAb+

## Association between Infection and Neutropenia/Lymphopenia

To evaluate the association between infection and neutropenia and also between infection and lymphopenia, the frequency of infections will be provided by the worst Common Terminology Criteria for Adverse Events (CTCAE) grades of neutropenia and lymphopenia, respectively. Infection outcomes considered for this analysis are any treatment-emergent infection, serious infection, and herpes zoster. For this analysis, no statistical comparison will be provided.

In addition, a summary table will be provided for treatment-emergent infections that were preceded or accompanied by neutropenia/lymphopenia. For this analysis, neutropenia is defined as CTCAE Grade 2 or greater. Infection events with onset date ≤14 days before or after the Grade 2 neutrophil/lymphocyte count collection date will be considered as infections preceded or accompanied by neutropenia.

## 4.6.3.2. Systemic Hypersensitivity Reactions (including cytokine release syndrome)

A search will be performed using the current MedDRA version Standardised MedDRA Queries (SMQs) to search for relevant events, using the following queries:

- Anaphylactic reaction SMQ (20000021)
- Hypersensitivity SMQ (20000214)
- Angioedema SMQ (20000024)

Events that satisfy the queries will be listed, by temporal order within patient ID, and will include SOC, PT, SMQ event categorization including detail on the scope (narrow or broad), reported AE term, AE onset and end dates, severity, seriousness, outcome, etc.

#### 4.6.3.3. Malignancies

Malignancies will be identified using terms from the malignant tumors SMQ (SMQ 20000194). Malignancies excluding nonmelanoma skin cancers (NMSC) and NMSC will be reported separately.

A listing including all malignancy cases will be provided. An NMSC flag will be provided using the following MedDRA PTs (the list will be updated depending on the MedDRA version used for analysis):

- Squamous cell carcinoma of skin (10041834)
- Bowen's disease (10006059)
- Basal cell carcinoma (10004146)
- Basosquamous carcinoma (10004178)
- Basosquamous carcinoma of skin (10004179)
- Squamous cell carcinoma (10041823)
- Skin squamous cell carcinoma metastatic (10077314)
- Skin cancer (10040808)
- Carcinoma in situ of skin (10007390)

The number and percentage of patients with TEAE-associated malignancies excluding NMSC and NMSC will be summarized by treatment group. In addition, the IR (for detail, see Section 4.6) and 95% CI will be calculated for the overall observation time. All cases identified by malignant tumors SMQ will be assessed after database lock by the medical team to determine (1) confirmed NMSC cases and (2) symptom and date that triggered the malignancy investigation or diagnosis. An additional listing based on medical review may also be provided if deemed necessary. All cases reported in the study database or by Lilly Safety System (LSS) report, disregarding the length of gap between the last treatment dose date and the event date will be included.

#### 4.6.3.4. Gastrointestinal Perforations

Treatment-emergent adverse events potentially related to gastrointestinal (GI) perforations will be analyzed using reported AEs. Identification of these events will be based on the PTs of the MedDRA Gastrointestinal Perforations SMQ (SMQ 20000107); note that this SMQ holds only narrow terms and has no broad terms. Potential GI perforations identified by the above SMQ search will be provided as a listing for internal review by the medical safety team. Each case will be assessed to determine whether it is a GI perforation. Frequency and relative frequency for each PT will be provided, ordered by decreasing frequency in the LY3471851 1800 $\mu$ g treatment group. Comparisons between each LY3471851 treatment group and placebo will be made using Fisher's exact test.

#### 4.6.4. Injection Site Reaction

If a participant spontaneously reports symptoms of an injection site reaction, an authorized member of the site staff who, in the opinion of the investigator, is qualified to assess reports of potential ISRs and who is not involved with any other study procedure will evaluate the participant's report.

The number and percentage of patients who experienced ISR will be summarized by treatment group and by visit. The number and percentage of patients with the following ISR records will be summarized by treatment group and by visit. Details about ISR records are referred to the Case Report Form (CRF).

- Anatomical location of the injection site reaction
- Abdomen Side
- Directionality of the anatomical location of the administration
- Arm side
- Whether the subject has any injection site erythema (reddening) or not
- Severity of the injection site erythema
- Whether the subject has any injection site induration (hardening or thickening of tissue) or not
- Severity of the injection site induration
- Whether the subject has any injection site pain (including burning) or not
- Severity of the injection site pain
- Whether the subject has any injection site pruritus
- Severity of the injection site pruritus

- Whether the subject has any injection site edema (swelling or accumulation of fluid in tissues at height above normal skin) or not
- Severity of the injection site edema
- When the Injection related event occurred in relationship to the study treatment

Ordinal logistic regression will be used for the ordinal ISR reported. The frequency of the maximum severity of ISRs will be summarized by treatment group.

### 4.6.5. Clinical Laboratory Evaluation

Laboratory evaluations will be summarized and analyzed for the following periods:

- Induction Period.
- Maintenance Period,
- Extension Period (including Extension Induction and Extension Maintenance)

All laboratory tests will be presented using the Système International of units (SI) and conventional (CN) units. For topics of safety in special groups and circumstances, laboratory test units will be specified for each analysis.

Lilly Large Clinical Trial Population Based (LCTPB) reference limits will be used to define the low and high limits because it is generally desirable for limits used for analyses to have greater specificity (identify fewer false positive cases) than reference limits used for individual patient management. When Lilly LCTPB reference ranges are unavailable, then central laboratory (Labcorp) reference ranges will be used. For the 4 key hepatic laboratory assessments (alanine aminotransferase [ALT], aspartate aminotransferase [AST], total bilirubin, and alkaline phosphatase [ALP]), central laboratory reference ranges (Labcorp) will be used and all results pertaining to these assessments will be included as a separate analysis to address the risk of liver injury as a special safety topic (see Section 4.6.3.1). Central laboratory reference ranges (Labcorp) will also be used to evaluate immunoglobulins and lymphocyte cell subsets (see Sections 4.6.5.2 and 4.6.5.6). See 6.10 for details of the reference range by laboratory analytes.

The low-density lipoprotein/high-density lipoprotein (LDL/HDL) ratio will be derived as the ratio of LDL cholesterol to HDL cholesterol. There are no Lilly LCTPB reference ranges or central lab reference ranges for the LDL/HDL ratio.

The following will be conducted for laboratory analyte measurements collected quantitatively:

• Box plots for observed values: Values at each visit (starting at randomization) and change from baseline to each visit and to last postbaseline measure will be displayed in box plots for patients who have a baseline and at least 1 postbaseline visit. For visits included in the treatment period, patients will be included only if the visit occurs on or before the date of treatment discontinuation/completion. Follow-up visit will be the first visit that occurred during the Follow-up period. Individual measurements outside of reference limits will also be displayed using distinct symbols overlaying the box plot. Original-scale data will be used for the display but for some analytes (e.g., immunoglobulins) a logarithmic scale will be used to aid in viewing the measures of central tendency and dispersion. Unplanned measurements will be excluded. Descriptive summary statistics will be included in a table below the box plot. These box plots will be

- used to evaluate trends over time and to assess a potential impact of outliers on central tendency summaries. A p-value for change from baseline to endpoint will be provided using an ANCOVA model with explanatory term for treatment and the baseline value as a covariate. Endpoint will be the last observation where patient is on treatment.
- Treatment-emergent high/low analyses: The number and percentage of patients with treatment-emergent high and low laboratory results at any time will be summarized by treatment group. Planned and unplanned measurements will be included. A treatment-emergent **high** result is defined as a change from a value less than or equal to the high limit at all baseline visits to a value greater than the high limit at any time during the treatment period and up to 60 days after treatment discontinuation. A treatment-emergent **low** result is defined as a change from a value greater than or equal to the low limit at all baseline visits to a value less than the low limit at any time during the treatment period and up to 60 days after treatment discontinuation. The Fisher's exact test will be used for the treatment comparisons.

For laboratory analyte measurements collected qualitatively, a listing of abnormal findings will be created. The listing will include patient ID, treatment group, laboratory collection date, analyte name, and analyte finding.

## 4.6.5.1. Abnormal Hepatic Tests

Analyses for abnormal hepatic tests involve 4 laboratory analytes: ALT, AST, total bilirubin, and ALP. Analyses for the change from baseline to last visit that occurred on or before the date of treatment discontinuation and shift tables are described in Section 4.6.5. This section describes additional analyses for the topic. The central laboratory reference ranges (Labcorp) will be used for ALT, AST, total bilirubin, and ALP hepatic laboratory assessments.

The number and percentage of patients with the following abnormal elevations in hepatic laboratory tests at any time up to 60 days after treatment discontinuation will be summarized by treatment group. LY3471851 groups will be compared to placebo using Fisher's exact text:

- The percentages of patients with an ALT measurement ≥3×, 5×, and 10× the central laboratory upper limit of normal (ULN) during the treatment and follow-up periods will be summarized for all patients with a postbaseline value.
- The percentages of patients with an AST measurement  $\ge 3 \times$ ,  $5 \times$ , and  $10 \times$  the central laboratory ULN during the treatment and follow-up periods will be summarized for all patients with a postbaseline value.
- The percentages of patients with a total bilirubin measurement  $\ge 2 \times$  the central laboratory ULN during the treatment period will be summarized for all patients with a postbaseline value.
- The percentages of patients with an ALP measurement  $\ge 3 \times$  the central laboratory ULN during the treatment and follow-up periods will be summarized for all patients with a postbaseline value.
Second, to further evaluate potential hepatotoxicity, an Evaluation of Drug-Induced Serious Hepatotoxicity (eDISH) plot will be created for all patients whether treated with LY3471851 and/or other treatment using the whole study and follow-up periods. Each patient with at least 1 postbaseline ALT and total bilirubin will be included in the eDISH. The points correspond to maximum total bilirubin and maximum ALT, even if not obtained from the same blood draw. A listing of patients potentially meeting Hy's rule will be provided (defined as greater than or equal to 3× ULN for ALT or AST, and greater than or equal to 2× ULN for total bilirubin, not necessarily at the same time).

Third, a listing will be provided to the medical safety team for internal review according to the following SMQs:

- Broad and narrow terms in the Liver-related investigations, signs and symptoms SMQ (SMQ 20000008)
- Broad and narrow terms in the Cholestasis and jaundice of hepatic origin SMQ (SMQ 20000009)
- Broad and narrow terms in the Hepatitis non-infectious SMQ (SMQ 20000010)
- Broad and narrow terms in the Hepatic failure, fibrosis and cirrhosis and other liver damage-related conditions SMQ (SMQ 20000013)
- Narrow terms in the Liver-related coagulation and bleeding disturbances SMQ (SMQ 20000015).

#### 4.6.5.2. Lymphocyte Subset Cell Counts

The following lymphocyte subsets will be analyzed:

CD3+ T Cells - %

CD3+ T Cells – Absolute

CD3+CD8+ T cells (CD8) – %

CD3+CD8+ T cells (CD8) – Absolute

CD3+CD4+ T cells (CD4) - %

CD3+CD4+ T cells (CD4) – Absolute

CD56+/CD16+ NK cells - %

CD56+/CD16+ NK cells – Absolute

CD19+ B cells – %

CD19+ B cells – Absolute

CD4/CD8 Ratio - Calculated

CD3+4+8+ %

CD3+4+8+ Abs

CD3/CD19 Ratio - Calculated

For each type of cells, both the absolute count and the relative count (i.e., as a percentage of the total lymphocyte population) will be analyzed. In addition, the ratio of CD4 cell counts to CD8 cell counts will be analyzed.

The analyses for these parameters will be performed using the same approaches as described for analysis of clinical laboratory measurements in Section 4.6.5. For determining treatment-emergent abnormal, high, or low lymphocyte subset cell counts, central laboratory reference ranges (Labcorp) will be used when available; note that reference ranges are available only for some of the lymphocyte subset cell count analytes.

## 4.6.5.3. Lipids Effects

Analyses for the change from baseline to last observation, and shift tables in total cholesterol, LDL cholesterol, HDL cholesterol, and triglycerides are described in Section 4.6.5.

Treatment-emergent adverse events potentially related to hyperlipidemia will also be analyzed, based on reported AEs. The target surveillance term "Hyperlipidemia" is a Lilly-defined MedDRA search criteria list that is a subset of the PTs in the MedDRA SMQ "Dyslipidemia" that are related to elevated or increased lipids. MedDRA PTs, each with a narrow scope from the SMQ, for the target surveillance term are shown in 6.9. Frequency and relative frequency for each PT will be provided, ordered by decreasing frequency in the LY3471851 1800µg treatment group.

#### 4.6.5.4. Renal Function Effects

Effects on renal function will be assessed through analyses of creatinine, which are described in Section 4.6.5.

#### 4.6.5.5. Elevations in Creatine Phosphokinase

Analyses of creatine phosphokinase are described in Section 4.6.5.

#### 4.6.5.6. Serum Immunoglobulin Concentrations

Each serum Ig concentration (IgA, IgG, and IgM) will be analyzed. The analyses for these parameters will be performed using the same approaches as described for analysis of clinical laboratory measurements in Section 4.6.5. For determining treatment-emergent abnormal, high, or low serum Ig concentrations for IgA, IgG, and IgM, central laboratory reference ranges (Labcorp) will be used.

## 4.6.6. Vital Signs and Other Physical Characteristics

Vital signs and physical characteristics include systolic blood pressure (SBP), diastolic blood pressure (DBP), pulse, weight, BMI, and body temperature. Original-scale data will be analyzed. When these parameters are analyzed as continuous numerical variables, unplanned measurements will be excluded. When these parameters are analyzed as categorical outcomes, planned and unplanned measurements will be included.

Vital signs and physical characteristics will be summarized and analyzed for the following periods:

• Induction Period

- Maintenance Period
- Extension Period

The planned analyses described for the laboratory analytes in Section 4.6.5 will be used to analyze the vital signs and physical characteristics.

Table KFAH.5 defines the low and high baseline values as well as the criteria used to define treatment-emergence based on postbaseline values. Postbaseline values include all values after baseline in the treatment and follow-up periods. The blood pressure and pulse rate criteria are consistent with the document *Selected Reference Limits for Blood Pressure, Orthostasis, and ECG Numerical Parameters (Including Heart Rate) for Use in Phase II-IV Clinical Trials Version 1.1* approved on 8 March 2013 as recommended by the Lilly Cardiovascular Safety Advisory Committee (CVSAC).

Table KFAH.5. Categorical Criteria for Abnormal Treatment-Emergent Blood Pressure and Pulse Measurement, and Categorical Criteria for Weight Changes for Adults

| | Low | High |
|---|---|---|
| Systolic Blood | ≤90 (low limit) and decrease from | ≥140 (high limit) and increase from highest |
| Pressure (mm Hg) | lowest value during baseline ≥20 if | value during baseline ≥20 if <140 at each |
| | >90 at each baseline visit | baseline visit |
| Diastolic Blood | ≤50 (low limit) and decrease from | ≥90 (high limit) and increase from highest |
| Pressure (mm Hg) | lowest value during baseline ≥10 if | value during baseline ≥10 if <90 at each |
| | >50 at each baseline visit | baseline visit |
| Pulse | <50 (low limit) and decrease from | >100 (high limit) and increase from highest |
| (beats per minute) | lowest value during baseline ≥15 if | value during baseline ≥15 if ≤100 at each |
| | ≥50 at each baseline visit | baseline visit |
| Weight | (Loss) decrease ≥7% from lowest | (Gain) increase ≥7% from highest value |
| (kilograms) | value during baseline | during baseline |

Abbreviation: mm Hg = millimeters of mercury.

## 4.6.7. Electrocardiograms

Detailed Electrocardiogram results are part of the clinical database for this study. Should an ECG be performed in association with an AE or medical history event, the occurrence of the ECG ("Yes/No") will be provided in a by-patient listing.

If any clinically significant ECG measurement occurs, this will be recorded as an AE. ECG data will not be analyzed.







#### 4.6.9. Suicidal Ideation/Behavior and Depression

During the study, suicidal ideation and behavior, and depression will be assessed prospectively by the investigator via signs and symptoms and through the use of the Columbia-Suicide Severity Rating Scale (C-SSRS) and the Quick Inventory of Depressive Symptomatology Self Report (QIDS-SR16).

Analyses will include:

- C-SSRS: Only a listing of the C-SSRS data will be provided.
- QIDS-SR16: Shift table will be provided showing the number and percentage of patients within each baseline category (maximum value) versus each post-baseline category (maximum value) by treatment. Additionally, outcomes such as any increase in depression will be compared between treatments.

## 4.7. Other Analyses

#### 4.7.1. Efficacy Subgroup Analysis

Subgroup analyses will be conducted on the mITT population for the following:

- Clinical remission
- Clinical response
- Endoscopic remission
- Endoscopic response
- Symptomatic remission
- Symptomatic response
- Histologic remission
- Histologic-endoscopic mucosal healing

The following subgroups (but not limited to only these) will be evaluated:

- Gender
- Age category
- Body weight
- Race
- Geographic region
- Baseline disease severity and activity
- Duration and location of disease

- Previous systemic therapy
- Previous advanced therapy, and
- Concomitant therapy for UC.

Descriptive statistics will be provided for each treatment and stratum of a subgroup as outlined, regardless sample size.

Each categorical variable will be analyzed individually with a logistic regression model that contains the treatment, the subgroup variable, and subgroup by treatment interaction. The treatment-by-subgroup interaction will be tested at the 10% significant level. Within each subgroup category, the proportion of responders by treatment, treatment differences, and 95% CIs will be displayed.

For continuous variables, MMRM analysis will be performed with subgroup-by-treatment interaction. Within each subgroup, LS means by treatment, LS mean differences, and 95% CIs will be displayed.

If the number of patients in any subgroup category is less than 10% of the total population, only summaries of the efficacy data will be provided. Additional subgroup analyses may be performed as deemed necessary.

## 4.7.2. Safety Subgroup Analyses

Safety subgroup analysis for safety related endpoints will be performed within the context of the integrated safety analysis. No safety subgroup analysis will be performed specifically for this study unless there is a potentially relevant finding during the periodic study safety reviews.

# 4.8. Interim Analyses

Analyses for the primary database lock will be conducted when all participants have completed the Induction Period (that is, have completed the Week 12 visit) or else have discontinued study treatment.

The following interim analyses may be conducted to assess the primary efficacy results:

- for early termination assessment and decision when approximately 50 patients have either completed the dosing induction period or discontinued study treatment,
- for early termination or Stage 2 dose decisions when approximately 100 patients have either completed the dosing induction period or discontinued study treatment,
- for early trigger to Phase 3 assessment when approximately 150 patients have either completed the dosing induction period or discontinued study treatment, and
- for Phase 3 study trigger when approximately 200 patients have either completed the dosing induction period or discontinued study treatment.

Bayesian pairwise comparisons (LY3471851 dose to placebo) will be employed for potential decisions at each interim analysis using Bayesian posterior probability. Note that Stage 2 treatment doses will be determined based on results of the second interim analysis and recommendations of the sponsor's IAC.

The interim efficacy results will be used for internal decision making to terminate or trigger planning activities associated with the investigational product and to aid development of PK/PD modeling. Hence, there will be no alpha adjustment at the interim analyses. For each pairwise comparison at each interim analysis, a alpha of 0.05 will be used. The study may not be stopped for positive efficacy. The assessment will be conducted by a sponsor assessment committee with a limited number of pre-identified team members who do not have direct site contact or data entry/validation responsibilities. To minimize any bias being introduced into the analysis of the study results, the SAP and PK/PD analysis plan will be finalized and approved before the first efficacy interim analysis is initiated.

Information that may unblind the study during the analyses will not be reported to study sites or the blinded study team until a decision is made to unblind the entire study team.

Ongoing monitoring of safety data (including AEs, SAEs, and selected laboratory measurements) will be continued throughout the study using blinded data. Reviewing details are specified in the trial level safety review (TLSR) plan or a separate document.

## **4.8.1.** Data Monitoring Committee (DMC)

Not applicable. An assessment of unblinded interim data will be conducted by an internal assessment committee (IAC) with a limited number of prespecified team members who do not have direct site contact or data entry or validation responsibilities. An AC charter will provide details on AC membership and the governing processes.

## 4.9. Changes to Protocol-Planned Analyses

Protocol deviations will be identified throughout the study. Important protocol deviations (IPDs) are defined as those deviations from the protocol that would potentially compromise patients' safety, data integrity, or study outcome.

A separate document known as the "The KFAH Trial Issues Management Plan" describes the categories and subcategories of important protocol deviations, whether or not these deviations are IPDPPs, and how the IPDs would be identified.

The number and percentage of patients having IPDs will be summarized within category and subcategory of deviations by dosing regimen for the mITT population.

## 5. Sample Size Determination

Approximately 200 participants, in total, may be randomized across all study stages.

During Stage 1, approximately 100 participants will be randomized to a high dose (CC μg) of LY3471851, a lower (CC μg) dose of LY3471851, or placebo groups in a 2:2:1 ratio.

During Stage 2, up to approximately 100 additional participants will be randomized. Stage 2 will have a placebo group and may have more LY3471851 treatment groups than Stage 1, or fewer, based on decisions taken after the last interim analysis of Stage 1.

The power calculations for this study assume the following:

- At end of study, three non-placebo treatment groups will have sample size of approximately either 40, 60, or 80 patients.
- At end of study, the placebo group will have a sample size of approximately 40 patients.
- For the sake of simplicity in the power calculation, it is assumed that there is no difference in treatment effect between advanced therapy-failed and conventional-failed patients. To simplify, it is also assumed that all treatment groups have the same treatment effect.
- It is assumed that the true placebo response rate is approximately 5% and the true treatment response is approximately 35%.
- Power is calculated for 3 hypothesis tests, 1 for each treatment group against placebo, and adjust for multiple comparisons using the conservative Bonferroni adjustment. Power is calculated using a family-wise error rate of  $\alpha$ =.05.

Given these assumptions, the power to reject the null hypotheses for the treatment groups with sample sizes equal to 40, 60, and 80 are 89.5%, 94.5%, and 96.5%, respectively. As an example, in a fixed design, with the placebo and LY3471851 treatment groups each having 80 participants, a 17% or larger difference between the groups can be detected with 90% power and assuming a 5% placebo effect.

## 6. Supporting Documentation

# 6.1. Appendix 1: Demographic and Baseline Characteristics

The patient's year of birth, sex, weight, height, smoking habits, previous biologic treatment, and other demographic characteristics are collected at the screening visit. Age and body mass index will be calculated.

Only the year of birth is collected at screening. For the purpose of age calculation, the month and day of birth will be imputed as July 01, of the year of birth. Age is computed as follows;

Age= (Informed Consent Date -Date of Birth +1)/365.25.

Demographic and baseline characteristics (including age, gender, race, and ethnicity) will be summarized for each treatment group.

Certain characteristics, that are collected at baseline or after baseline but not summarized in the demographic summary, will be reported as a listing.

No inferential analysis for the comparability of baseline covariates across treatment groups will be performed.

## **6.2.** Appendix 2: Preexisting Conditions

Preexisting condition is defined the condition/event recorded on the Preexisting Conditions and Medical History electronic case report form (eCRF) page with a start date prior to the date of informed consent, and no end date (that is, the event is ongoing) or an end date on or after the date of informed consent. In addition, the AEs occurring prior to first dose are also included. Notice if a preexisting condition worsens in severity on or after the date of informed consent, it will be recorded as an AE on the AE eCRF page with the date of worsening as the start date. The number and percentage of patients with preexisting conditions will be summarized by treatment group using the MedDRA Preferred Term (PT) nested within System Organ Class (SOC). Summaries will be performed for the ITT population.

# **6.3.** Appendix 3: Treatment Compliance

Study treatment administration and compliance will be listed for all entered patients. The number and percentage of patients who are treatment compliant by week (that is, at each injection time point) will be summarized by treatment group for each treatment period.

No patient will be excluded from the ITT population as a consequence of significant noncompliance.

Participants who are noncompliant with treatment will be listed by treatment group.

No analyses are planned to assess treatment compliance.

# 6.4. Appendix 4: Prior and Concomitant Therapy

Prior and concomitant medications will be summarized by treatment group and will be classified into anatomical therapeutic chemical (ATC) drug classes using the latest version of the World Health Organization (WHO) drug dictionary. Medication start and stop dates will be compared to

the date of first dose of treatment in each treatment period to allow medications to be classified as Concomitant for each treatment period.

Prior medications are those medications that start and stop prior to the date of first dose of study treatment. Concomitant medications are those medications that start before, on or after the first day of study treatment of the defined treatment period and continue into the treatment period.

## 6.5. Appendix 5: Clinical Trial Registry Analyses

Additional analyses will be performed for the purpose of fulfilling the Clinical Trial Registry (CTR) requirements.

Analyses provided for the CTR requirements include the following:

Summary of adverse events, provided as a dataset which will be converted to an XML file. Both Serious Adverse Events and 'Other' Adverse Events are summarized: by treatment group, by MedDRA preferred term.

- An adverse event is considered 'Serious' whether or not it is a treatment emergent adverse event (TEAE).
- An adverse event is considered in the 'Other' category if it is both a TEAE and is not serious. For each Serious AE and 'Other' AE, for each term and treatment group, the following are provided:
  - o the number of participants at risk of an event
  - o the number of participants who experienced each event term
  - o the number of events experienced.
- Consistent with www.ClinicalTrials.gov requirements, 'Other' AEs that occur in fewer than 5% of patients/subjects in every treatment group may not be included if a 5% threshold is chosen (5% is the minimum threshold).

AE reporting is consistent with other document disclosures for example, the CSR, manuscripts, and so forth.

# 6.6. Appendix 6: Daily Diary Calculations

Weekly summary measures of daily diary data will be created for each patient. The 7-day period associated with each week will be defined using a visit centric approach. The table below displays the interval for each week:

| Week (Visit) | Start Day <sup>a</sup> | End Day <sup>a</sup> |
|---|---|---|
| Baseline | Week 0 Visit Date – 7 | Week 0 Visit Date – 1 |
| Week 1 (V3) | Max(Week 0 Visit Date, Week 1 Visit Date – 7) | Week 1 Visit Date – 1 |
| Week 2 (V4) | Max(Week 1 Visit Date, Week 2 Visit Date – 7) | Week 2 Visit Date – 1 |

| Week 3 | Max (Week 2 Visit Date, Week 4 Visit Date – 14) | Week 4 Visit Date – 8 |
|---|---|---|
| Week 4 (V5) | Max (Week 2 Visit Date, Week 4 Visit Date – 7) | Week 4 Visit Date – 1 |
| Week 5 | Max (Week 4 Visit Date, Week 6 Visit Date – 14) | Week 6 Visit Date – 8 |
| Week 6 (V6) | Max (Week 4 Visit Date, Week 6 Visit Date – 7) | Week 6 Visit Date – 1 |
| Week 7 | Max (Week 6 Visit Date, Week 8 Visit Date – 14) | Week 8 Visit Date – 8 |
| Week 8 (V7) | Max (Week 6 Visit Date, Week 8 Visit Date – 7) | Week 8 Visit Date – 1 |
| Week 9 | Max (Week 8 Visit Date, Week 10 Visit Date – 14) | Week 10 Visit Date – 8 |
| Week 10 (V8) | Max (Week 8 Visit Date, Week 10 Visit Date – 7) | Week 10 Visit Date – 1 |
| Week 11 | Max (Week 10 Visit Date, Week 12 Visit Date – 14) | Week 12 Visit Date – 8 |
| Week 12 (V9) | Max (Week 10 Visit Date, Week 12 Visit Date – 7) | Week 12 Visit Date – 1 |
| Week 13 | Max (Week 12 Visit Date, Week 14 Visit Date – 14) | Week 14 Visit Date – 8 |
| Week 14 (V10) | Max (Week 12 Visit Date, Week 14 Visit Date – 7) | Week 14 Visit Date – 1 |
| Week 15 | Max (Week 14 Visit Date, Week 16 Visit Date – 14) | Week 16 Visit Date – 8 |
| Week 16 (V11) | Max (Week 14 Visit Date, Week 16 Visit Date – 7) | Week 16 Visit Date – 1 |
| Week 17 | Max (Week 16 Visit Date, Week 18 Visit Date – 14) | Week 18 Visit Date – 8 |
| Week 18 (V12) | Max (Week 16 Visit Date, Week 18 Visit Date – 7) | Week 18 Visit Date – 1 |
| Week 19 | Max (Week 18 Visit Date, Week 20 Visit Date – 14) | Week 20 Visit Date – 8 |
| Week 20 (V13) | Max (Week 18 Visit Date, Week 20 Visit Date – 7) | Week 20 Visit Date – 1 |
| Week 21 | Max (Week 20 Visit Date, Week 22 Visit Date – 14) | Week 22 Visit Date – 8 |
| Week 22 (V14) | Max (Week 20 Visit Date, Week 22 Visit Date – 7) | Week 22 Visit Date – 1 |
| Week 23 | Max (Week 22 Visit Date, Week 24 Visit Date – 14) | Week 24 Visit Date – 8 |
| Week 24 (V15) | Max (Week 22 Visit Date, Week 24 Visit Date – 7) | Week 24 Visit Date – 1 |
| Week 25 | Max (Week 24 Visit Date, Week 26 Visit Date – 14) | Week 26 Visit Date – 8 |
| Week 26 (V16) | Max (Week 24 Visit Date, Week 26 Visit Date – 7) | Week 26 Visit Date – 1 |
| Week 27 | Max(Week 26 Visit Date, Week 28 Visit Date – 14) | Week 28 Visit Date – 1 |
| Week 28 (V17) | Max(Week 26 Visit Date, Week 28 Visit Date – 7) | Week 28 Visit Date – 1 |

| Week 29 | Max (Week 28 Visit Date, Week 30 Visit Date – 14) | Week 30 Visit Date – 8 |
|---|---|---|
| Week 30 (V18) | Max (Week 28 Visit Date, Week 30 Visit Date – 7) | Week 30 Visit Date – 1 |
| Week 31 | Max (Week 30 Visit Date, Week 32 Visit Date – 14) | Week 32 Visit Date – 8 |
| Week 32 (V19) | Max (Week 30 Visit Date, Week 32 Visit Date – 7) | Week 32 Visit Date – 1 |
| Week 33 | Max (Week 32 Visit Date, Week 34 Visit Date – 14) | Week 34 Visit Date – 8 |
| Week 34 (V20) | Max (Week 32 Visit Date, Week 34 Visit Date – 7) | Week 34 Visit Date – 1 |
| Week 35 | Max (Week 34 Visit Date, Week 36 Visit Date – 14) | Week 36 Visit Date – 8 |
| Week 36 (V21) | Max (Week 34 Visit Date, Week 36 Visit Date – 7) | Week 36 Visit Date – 1 |
| Week 37 | Max (Week 36 Visit Date, Week 38 Visit Date – 14) | Week 38 Visit Date – 8 |
| Week 38 (V22) | Max (Week 36 Visit Date, Week 38 Visit Date – 7) | Week 38 Visit Date – 1 |
| Week 39 | Max (Week 38 Visit Date, Week 40 Visit Date – 14) | Week 40 Visit Date – 8 |
| Week 40 (V23) | Max (Week 38 Visit Date, Week 40 Visit Date – 7) | Week 40 Visit Date – 1 |
| Week 41 | Max (Week 40 Visit Date, Week 42 Visit Date – 14) | Week 42 Visit Date – 8 |
| Week 42 (V24) | Max (Week 40 Visit Date, Week 42 Visit Date – 7) | Week 42 Visit Date – 1 |
| Week 43 | Max (Week 42 Visit Date, Week 44 Visit Date – 14) | Week 44 Visit Date – 8 |
| Week 44 (V25) | Max (Week 42 Visit Date, Week 44 Visit Date – 7) | Week 44 Visit Date – 1 |
| Week 45 | Max (Week 44 Visit Date, Week 46 Visit Date – 14) | Week 46 Visit Date – 8 |
| Week 46 (V26) | Max (Week 44 Visit Date, Week 46 Visit Date – 7) | Week 46 Visit Date – 1 |
| Week 47 | Max (Week 46 Visit Date, Week 48 Visit Date – 14) | Week 48 Visit Date – 8 |
| Week 48 (V27) | Max (Week 46 Visit Date, Week 48 Visit Date – 7) | Week 48 Visit Date – 1 |
| Week 49 | Max (Week 48 Visit Date, Week 50 Visit Date – 14) | Week 50 Visit Date – 8 |
| Week 50 (V28) | Max (Week 48 Visit Date, Week 50 Visit Date – 7) | Week 50 Visit Date – 1 |
| Week 51 | Max (Week 50 Visit Date, Week 52 Visit Date – 14) | Week 52 Visit Date – 8 |
| Week 52 (V29) | Max (Week 50 Visit Date, Week 52 Visit Date – 7) | Week 52 Visit Date – 1 |

Abbreviations: V = Visit.

<sup>a</sup> If End Day < Start Day, do not assign specified visit week. Visit date will be calculated by selecting the first date from the following list (i.e., first in list order): (1) date of earliest bowel preparation if bowel preparation date is available, (2) date of endoscopy if endoscopy was performed, (3) date of treatment if treatment was given, (4) office visit date if available, or (5) imputed date of visit center of the protocol-defined window for that visit. The screening endoscopy is assumed to be associated with the Week 0 visit.

For the Mayo SF and RB subscores, the most recent 3 nonmissing days of the 7-day period in the table above will be averaged and rounded to the nearest integer to calculate the weekly score for each patient. Patients with less than 3 measurements in the 7 day period will be considered missing.

For the Bristol Stool Scale the worst (i.e. maximum) of the available measures during the 7 period in the table above will be used to calculate a weekly score for each patient. If fewer than 4 days are available (i.e., not missing), the patient will be considered to be missing data for that week.

For all other daily diary measures, all available days of the 7 days will be averaged and rounded to the nearest integer to calculate the weekly score for each patient. If fewer than 4 days are available (i.e., not missing), the patient will be considered to be missing data for that week.

If multiple diary assessments on a single day are present, use the earliest nonmissing assessment. Data from the following days will be considered missing: (i) days when patients receive bowel preparation, (ii) the day of an endoscopy, and (iii) two days after an endoscopy.

If the baseline assessment is missing per the above rules, the first available postbaseline assessment starting with Week 1 will be used to impute the baseline so that the patient can be included in the analysis.

# 6.7. Appendix 7: Execution for Bayesian Model Averaging

#### 6.7.1. R DREAMER Package to Execute BMA

BMA will be executed using the R package *DREAMER*: **D**ose **RE**sponse b**A**yesian **M**odel averaging. *DREAMER* package and supporting documentation may be found at <u>GitHub - rich-payne/dreamer</u> and on CRAN.

#### 6.7.2. BMA Components, Priors, and Weights

E-max, quadratic, log-quadratic, linear, and log-linear dose response models are the prespecified component to the BMA model that will be used to analyze the KFAH dose response and are described in the DREAMER supporting documentation. BMA components and weights are summarized in **** The priors for each parameter are normal distributions, except  $b_4$  in the Sigmoidal EMAX model, which is truncated normal (to be positive). A logistic link function will be used for each model.

Table KFAH.6. Prespecified Dose Response Models with Prior

| Component | Weight | Model | Parameter | mu | sigma |
|---|---|---|---|---|---|
| Sigmoidal EMAX | 1/6 | $(b_2 - b_1)d^{b_4}$ | $b_I$ | -2 | 2 |
| | | $f(d) = b_1 + \frac{(b_2 - b_1)a}{\exp(b_3 b_4) + d^{b_4}}$ | $b_2$ | 0 | 4 |

| | | | $b_3$ | log(CCI | log(600) |
|---|---|---|---|---|---|
| | | | $b_4$ | 1 | 2 |
| Hyperbolic EMAX | 1/6 | $f(d) = b_1 + \frac{(b_2 - b_1)d}{\exp(b_3) + d}$ | $b_{I}$ | -2 | 2 |
| | | $f(a) = b_1 + \frac{1}{\exp(b_3) + d}$ | $b_2$ | 0 | 4 |
| | | | $b_3$ | log(CCI | log(600) |
| Quadratic | 1/6 | $f(d) = b_1 + b_2 d + b_3 d^2$ | $b_1$ | -2 | 2 |
| | | | $b_2$ | 0 | 2 |
| | | | $b_3$ | 0 | 2 |
| Log-Quadratic | 1/6 | $f(d) = b_1 + b_2 \log(d+1)$ | $b_1$ | -2 | 2 |
| | | $+ b_3 \log(d+1)^2$ | $b_2$ | 0 | 1 |
| | | | $b_3$ | 0 | 1 |
| Linear | 1/6 | $f(d) = b_1 + b_2 d$ | $b_1$ | -2 | 2 |
| | | | $b_2$ | 0 | 2 |
| Log-Linear | 1/6 | $f(d) = b_1 + b_2 \log(d+1)$ | $b_1$ | -2 | 2 |
| | | | $b_2$ | 0 | 1 |

6.8. Appendix 8: List of MedDRA Preferred Terms for Potential Opportunistic Infections (POI)

| Category | Potential | Preferred Term | Preferred Term | Lilly Defined |
|---|---|---|---|---|
| | Opportunistic | (MedDRA Version | Code | Classification |
| | Infection | 22.1) | | |
| Mycobacterial/ | Nocardiosis (II) | Nocardia sepsis | 10064952 | Narrow |
| Actino | | Nocardiosis | 10029444 | |
| | | Nocardia test positive | 10070131 | Broad |
| Mycobacterial/<br>Actino | Nontuberculous mycobacterium | Atypical mycobacterial infection | 10061663 | Narrow |
| | disease (II) | Atypical mycobacterial lower respiratory tract infection | 10075026 | |
| | | Atypical mycobacterial lymphadenitis | 10003755 | |
| | | Atypical mycobacterium pericarditis | 10055036 | |
| | | Atypical mycobacterial pneumonia | 10071075 | |
| | | Borderline leprosy | 10006029 | |
| | | Bovine tuberculosis | 10006049 | |
| | | Indeterminate leprosy | 10021700 | |
| | | Leprosy | 10024229 | |
| | | Lepromatous leprosy | 10024227 | |
| | | Mycobacterial infection | 10062207 | |
| | | Mycobacterial peritonitis | 10073514 | |

| Category | Potential<br>Opportunistic<br>Infection | Preferred Term<br>(MedDRA Version<br>22.1) | Preferred Term<br>Code | Lilly Defined<br>Classification |
|---|---|---|---|---|
| | | Mycobacterium abscessus infection | 10064789 | |
| | | Mycobacterium avium complex immune restoration disease | 10058449 | |
| | | Mycobacterium avium complex infection | 10058806 | |
| | | Mycobacterium chelonae infection | 10071401 | |
| | | Mycobacterium fortuitum infection | 10049659 | |
| | | Mycobacterium kansasii infection | 10028447 | |
| | | Mycobacterium<br>marinum infection | 10028452 | |
| | | Mycobacterium ulcerans infection | 10066289 | |
| | | Superinfection<br>mycobacterial | 10075381 | |
| | | Tuberculoid leprosy | 10044729 | |
| | | Type 1 lepra reaction | 10070516 | |
| | | Type 2 lepra reaction | 10070517 | |
| | | Atypical mycobacterium test positive | 10070326 | Broad |
| | | Mycobacterial disease carrier | 10075025 | |
| | | Mycobacterium leprae test positive | 10070324 | |
| | | Mycobacterium test | 10070407 | |
| | | Mycobacterium test positive | 10070323 | |
| | | Ureaplasmal ulvovaginitis | 10081280 | |
| Mycobacterial/<br>Actino | Tuberculosis (I) | Adrenal gland<br>tuberculosis | 10001358 | Narrow |
| | | Bone tuberculosis | 10056377 | |
| | | Choroid tubercles | 10008779 | |
| | | Congenital tuberculosis | 10010657 | |
| | | Conjunctivitis tuberculous | 10010754 | |
| | | Cutaneous tuberculosis | 10011684 | |
| | | Disseminated Bacillus<br>Calmette-Guerin | 10076666 | |
| | | infection | | |

| Category | Potential | Preferred Term | Preferred Term | Lilly Defined |
|---|---|---|---|---|
| | Opportunistic | (MedDRA Version | Code | Classification |
| | Infection | 22.1) | | |
| | | Disseminated | 10013453 | |
| | | tuberculosis | | |
| | | Ear tuberculosis | 10014027 | |
| | | Epididymitis | 10015004 | |
| | | tuberculous | | |
| | | Extrapulmonary | 10064445 | |
| | | tuberculosis | 10051150 | |
| | | Female genital tract | 10061150 | |
| | | tuberculosis | 10050505 | |
| | | Immune reconstitution | 10072797 | |
| | | inflammatory syndrome associated tuberculosis | | |
| | | | 10075269 | |
| | | Intestinal tuberculosis | 10075268 | $\dashv$ |
| | | Joint tuberculosis | 10056367 | _ |
| | | Lupus vulgaris | 10025143 | |
| | | Lymph node | 10025183 | |
| | | tuberculosis Mala capital tract | 10061234 | <del> </del> |
| | | Male genital tract tuberculosis | 10001234 | |
| | | Meningitis tuberculous | 10027259 | |
| | | Oesophageal | 10027239 | _ |
| | | tuberculosis | 10030200 | |
| | | Oral tuberculosis | 10076879 | |
| | | Pericarditis tuberculous | 10055069 | |
| | | Peritoneal tuberculosis | 10053583 | <del> </del> |
| | | | | _ |
| | | Prostatitis tuberculous | 10064743<br>10066927 | |
| | | Pulmonary tuberculoma | 10000927 | |
| | | Pulmonary tuberculosis | | |
| | | Renal tuberculosis | 10038534 | _ |
| | | Salpingitis tuberculous | 10039463 | |
| | | Silicotuberculosis | 10068876 | |
| | | Spleen tuberculosis | 10041640 | |
| | | Thyroid tuberculosis | 10043774 | _ |
| | | Tuberculoma of central | 10052883 | |
| | | nervous system | 1001155 | |
| | | Tuberculosis | 10044755 | |
| | | Tuberculosis bladder | 10044758 | _ |
| | | Tuberculosis | 10061390 | |
| | | gastrointestinal | 10050120 | $\dashv$ |
| | | Tuberculosis liver | 10058120 | $\dashv$ |
| | | Tuberculosis of central | 10061391 | |
| | | nervous system | 10044010 | _ |
| | | Tuberculosis of eye | 10044819 | |

| Category | Potential Opportunistic Infection | Preferred Term<br>(MedDRA Version<br>22.1) | Preferred Term<br>Code | Lilly Defined<br>Classification |
|---|---|---|---|---|
| | | Tuberculosis of genitourinary system | 10044828 | |
| | | Tuberculosis of intrathoracic lymph nodes | 10044846 | |
| | | Tuberculosis of peripheral lymph nodes | 10044965 | |
| | | Tuberculosis ureter | 10045026 | |
| | | Tuberculous abscess central nervous system | 10052884 | |
| | | Tuberculous endometritis | 10071559 | |
| | | Tuberculous laryngitis | 10045072 | |
| | | Tuberculous pleurisy | 10045104 | |
| | | Tuberculous<br>tenosynovitis | 10059161 | |
| | | Interferon gamma release assay | 10073542 | Broad |
| | | Interferon gamma release assay positive | 10072866 | |
| | | Mycobacterium<br>tuberculosis complex<br>test | 10070472 | |
| | | Mycobacterium<br>tuberculosis complex<br>test positive | 10070325 | |
| | | Tuberculid | 10044725 | |
| | | Tuberculin test | 10044726 | |
| | | Tuberculin test false negative | 10074840 | |
| | | Tuberculin test positive | 10044728 | |
| Bacteria | Bartonellosis | Bacillary angiomatosis | 10003971 | Narrow |
| | (disseminated disease | Trench fever | 10044582 | |
| | only) (V) | Bartonella test | 10075209 | Broad |
| | | Bartonella test positive | 10070157 | |
| | | Bartonellosis | 10004145 | |
| | | Cat scratch disease | 10007729 | |
| | | Peliosis hepatis | 10034229 | _ |
| | 0 11 | Splenic peliosis | 10068851 | NT. |
| | Campylobacteriosis | Campylobacter sepsis | 10070681 | Narrow |
| | (invasive disease only) (V) | Campylobacter colitis Campylobacter | 10076769<br>10007048 | Broad |
| | | gastroenteritis Campylobacter infection | 10051226 | |

| Category | Potential | Preferred Term | Preferred Term | Lilly Defined |
|---|---|---|---|---|
| <i>.</i> | Opportunistic | (MedDRA Version | Code | Classification |
| | Infection | 22.1) | | |
| | | Campylobacter test | 10070025 | |
| | | positive | | |
| | Legionellosis (II) | Legionella infection | 10061266 | Narrow |
| | | Pneumonia legionella | 10035718 | |
| | | Pontiac fever | 10054161 | |
| | | Legionella test | 10070410 | Broad |
| | | Legionella test positive | 10070092 | |
| Bacteria | Listeria | Listeria encephalitis | 10054116 | Narrow |
| | monocytogenes | Listeria sepsis | 10063085 | |
| | (invasive disease | Meningitis listeria | 10027248 | |
| | only) (II) | Listeria test | 10075707 | Broad |
| | | Listeria test positive | 10070094 | |
| | | Listeriosis | 10024641 | |
| | Salmonellosis | Aortitis salmonella | 10074937 | Narrow |
| | (invasive disease | Arthritis salmonella | 10003271 | |
| | only) (II) | Meningitis salmonella | 10027254 | |
| | | Osteomyelitis | 10031262 | |
| | | salmonella | | |
| | | Paratyphoid fever | 10033971 | |
| | | Pneumonia salmonella | 10035733 | |
| | | Salmonella bacteraemia | 10058924 | |
| | | Salmonella sepsis | 10058878 | |
| | | Typhoid fever | 10045275 | |
| | | Salmonella test positive | 10070127 | Broad |
| | | Salmonellosis | 10039447 | |
| | | Salmonella test | 10079854 | |
| Bacteria | Shigellosis (invasive | Shigella sepsis | 10074481 | Narrow |
| | disease only) (V) | Shigella infection | 10054178 | Broad |
| | • / ` / | Shigella test positive | 10070129 | |
| | Vibriosis (invasive | Gastroenteritis vibrio | 10017917 | Broad |
| | disease due to $V$ . | Vibrio test positive | 10070161 | |
| | vulnificus) (V) | None | | Narrow |
| | Infective Pneumonia | Pneumonia | 10079866 | |
| | SMQ | acinetobacter | | |
| | | Pneumonia proteus | 10079867 | Narrow |
| | | Pneumonia serratia | 10079868 | |
| Fungal | Aspergillosis | Aspergillosis oral | 10003489 | |
| 6 | (invasive disease | Cerebral aspergillosis | 10051597 | |
| | only) (II) | Meningitis aspergillus | 10073245 | |
| | • / ` / | Oro-pharyngeal | 10053029 | |
| | | aspergillosis | | |
| | | Aspergillus infection | 10074171 | |
| | | Aspergillus test | 10070450 | |
| | | Aspergillus test positive | 10070448 | |

| Category | Potential Opportunistic Infection | Preferred Term<br>(MedDRA Version<br>22.1) | Preferred Term<br>Code | Lilly Defined<br>Classification |
|---|---|---|---|---|
| | | Bronchopulmonary aspergillosis | 10006473 | |
| | | Sinusitis aspergillus | 10051016 | |
| | Blastomycosis (IV) | Blastomycosis | 10005098 | Narrow |
| | | Epididymitis<br>blastomyces | 10015001 | |
| | | Osteomyelitis<br>blastomyces | 10031255 | |
| | | Pneumonia blastomyces | 10035671 | |
| | | None | | Broad |
| | Candidiasis (invasive disease, or oral not | Candida<br>endophthalmitis | 10059449 | Narrow |
| | limited to the tongue) | Candida osteomyelitis | 10064699 | |
| | (II) | Candida pneumonia | 10053158 | |
| | | Candida retinitis | 10068612 | |
| | | Candida sepsis | 10053166 | |
| | | Candida urethritis | 10081262 | |
| | | Candidiasis of trachea | 10064459 | |
| | | Cerebral candidiasis | 10078126 | |
| | | Endocarditis candida | 10014669 | |
| | | Gastrointestinal candidiasis | 10017938 | |
| | | Hepatic candidiasis | 10040652 | |
| | | Hepatosplenic | 10049653<br>10051590 | |
| | | candidiasis | | |
| | | Meningitis candida | 10027205 | |
| | | Oesophageal candidiasis | 10030154 | |
| | | Oral candidiasis | 10030963 | |
| | | Oropharyngeal candidiasis | 10050346 | |
| | | Peritoneal candidiasis | 10056562 | |
| | | Splenic candidiasis | 10051725 | |
| | | Systemic candida | 10042938 | |
| | | Bladder candidiasis | 10058523 | Broad |
| | | Candida infection | 10074170 | |
| | | Candida test | 10070453 | |
| | | Candida test positive | 10070451 | |
| | | Mucocutaneous | 10028080 | |
| | | candidiasis <sup>1</sup> | | |
| | | Respiratory moniliasis | 10038705 | |
| | Coccidioidomycosis | Coccidioides | 10054214 | Narrow |
| | (II) | encephalitis | | |
| | | Coccidioidomycosis | 10009825 | |
| | | Cutaneous coccidioidomycosis | 10068747 | |

| Category | Potential<br>Opportunistic<br>Infection | Preferred Term<br>(MedDRA Version<br>22.1) | Preferred Term<br>Code | Lilly Defined<br>Classification |
|---|---|---|---|---|
| | | Meningitis coccidioides | 10027207 | |
| | | None | | Broad |
| | Cryptococcosis (II) | Cryptococcal cutaneous infection | 10054216 | Narrow |
| | | Cryptococcal fungaemia | 10067112 | |
| | | Cryptococcosis | 10011490 | |
| | | Disseminated cryptococcosis | 10013439 | |
| | | Gastroenteritis | 10011485 | |
| | | Cryptococcal Maningitis anymtococcal | 10027200 | |
| | | Meningitis cryptococcal | 10027209 | |
| | | Neurocryptococcosis Proumonia aruntagagas | 10068368 | |
| | | Pneumonia cryptococcal | 10067565<br>10070456 | Broad |
| | | Cryptococcus test Cryptococcus test positive | 10070455 | Broad |
| | Histoplasmosis (II) | Acute pulmonary histoplasmosis | 10001027 | Narrow |
| | | Chronic pulmonary histoplasmosis | 10009115 | |
| | | Endocarditis<br>histoplasma | 10014676 | |
| | | Histoplasmosis | 10020141 | |
| | | Histoplasmosis cutaneous | 10049142 | |
| | | Histoplasmosis<br>disseminated | 10020144 | |
| | | Meningitis histoplasma | 10027243 | |
| | | Pericarditis histoplasma | 10027243 | |
| | | Retinitis histoplasma | 10038912 | |
| | | Presumed ocular<br>histoplasmosis<br>syndrome | 10063664 | Broad |
| | Microsporidiosis (IV) | Microsporidia infection | 10053982 | Narrow |
| | | None | | Broad |
| | Other invasive fungi: | Allescheriosis | 10001754 | Narrow |
| | Mucormycosis | Fusarium infection | 10051919 | |
| | (=zygomycosis) | Mucormycosis | 10028098 | |
| | [Rhizopus, Mucor, | Scedosporium infection | 10059045 | |
| | and Lichtheimia], Scedosporum/ | Pseudallescheria infection | 10061919 | |
| | Pseudallescheria | Pseudallescheria sepsis | 10058973 | |
| | boydii, Fusarium (II) | See "Non-specific terms" below | | Broad |

| Category | Potential Opportunistic Infection | Preferred Term<br>(MedDRA Version<br>22.1) | Preferred Term<br>Code | Lilly Defined<br>Classification |
|---|---|---|---|---|
| | Paracoccidioides infections (V) | Paracoccidioides infection | 10061906 | Narrow |
| | infections (v) | None | | Broad |
| | Penicillium marneffei | Penicillium infection | 10078580 | Narrow |
| | (V) | | 100/8380 | |
| | | None | 10072756 | Broad |
| | Pneumocystis | Pneumocystis jirovecii | 10073756 | Narrow |
| | jirovecii (II) | infection | 10072755 | |
| | | Pneumocystis jirovecii | 10073755 | |
| | | pneumonia | 10069725 | Danad |
| | | Blood beta-D-glucan | 10068725<br>10051795 | Broad |
| | | Blood beta-D-glucan abnormal | 10051/95 | |
| | | | 10051793 | |
| | | Blood beta-D-glucan increased | 10031793 | |
| | | Gomori methenamine | 10075549 | |
| | | silver stain | 100/3349 | |
| | | Carbon monoxide | 10065906 | |
| | | diffusing capacity | 10003900 | |
| | | decreased | | |
| | | Carbon monoxide | 10071738 | |
| | | diffusing capacity | 100/1/38 | |
| | | Pneumocystis test | 10070454 | |
| | | positive | 10070434 | |
| | Sporothrix schenckii | Cutaneous | 10011676 | Narrow |
| | (V) | sporotrichosis | 10011070 | Narrow |
| | (*) | Sporotrichosis | 10041736 | |
| | | None | 10041730 | Broad |
| Viral | Cytomegalovirus | Cytomegalovirus | 10048843 | Narrow |
| VIIIII | disease (V) | chorioretinitis | 10040043 | Narrow |
| | discuse (1) | Cytomegalovirus colitis | 10048983 | |
| | | Cytomegalovirus | 10049014 | |
| | | duodenitis | 100.501. | |
| | | Cytomegalovirus | 10049074 | |
| | | enteritis | 100.507. | |
| | | Cytomegalovirus | 10049015 | |
| | | enterocolitis | | |
| | | Cytomegalovirus | 10049016 | |
| | | gastritis | | |
| | | Cytomegalovirus | 10051349 | |
| | | gastroenteritis | | |
| | | Cytomegalovirus | 10052817 | |
| | | gastrointestinal infection | | |
| | | Cytomegalovirus | 10075619 | |
| | | gastrointestinal ulcer | | |

| Category | Potential | Preferred Term | Preferred Term | Lilly Defined |
|---|---|---|---|---|
| | Opportunistic | (MedDRA Version | Code | Classification |
| | Infection | 22.1) | | |
| | | Cytomegalovirus | 10011830 | |
| | | hepatitis | | |
| | | Cytomegalovirus | 10011831 | |
| | | infection | | |
| | | Cytomegalovirus | 10011834 | |
| | | mononucleosis | | |
| | | Cytomegalovirus | 10065036 | |
| | | mucocutaneous ulcer | | |
| | | Cytomegalovirus | 10065621 | |
| | | myelomeningoradiculitis | | |
| | | Cytomegalovirus | 10056261 | |
| | | myocarditis | | |
| | | Cytomegalovirus | 10079095 | |
| | | nephritis | | |
| | | Cytomegalovirus | 10049018 | |
| | | oesophagitis | | |
| | | Cytomegalovirus | 10049566 | |
| | | pancreatitis | | |
| | | Cytomegalovirus | 10056721 | |
| | | pericarditis | | |
| | | Cytomegalovirus | 10056262 | |
| | | syndrome | | |
| | | Cytomegalovirus | 10051350 | |
| | | urinary tract infection | | |
| | | Cytomegalovirus | 10058854 | |
| | | viraemia | | |
| | | Disseminated | 10049075 | |
| | | cytomegaloviral | | |
| | | infection | | |
| | | Encephalitis | 10014586 | |
| | | cytomegalovirus | | |
| | | Pneumonia | 10035676 | |
| | | cytomegaloviral | | |
| | | Cytomegalovirus test | 10061806 | Broad |
| | | Cytomegalovirus test | 10051620 | |
| | | positive | | |
| | HBV reactivation | None | | Narrow |
| | (IV) | Asymptomatic viral | 10063838 | Broad |
| | | hepatitis | | |
| | | Chronic hepatitis B | 10008910 | |
| | | HBV-DNA polymerase | 10058937 | |
| | | increased | | |
| | | Hepatitis B | 10019731 | |
| | | Hepatitis B antigen | 10063414 | |

| Category | Potential Opportunistic Infection | Preferred Term<br>(MedDRA Version<br>22.1) | Preferred Term<br>Code | Lilly Defined<br>Classification |
|---|---|---|---|---|
| | | Hepatitis B antigen positive | 10063411 | |
| | | Hepatitis B core antigen | 10051160 | |
| | | Hepatitis B core antigen positive | 10052328 | |
| | | Hepatitis B DNA assay | 10060027 | |
| | | Hepatitis B DNA assay positive | 10060047 | |
| | | Hepatitis B DNA increased | 10068379 | |
| | | Hepatitis B e antigen | 10050914 | |
| | | Hepatitis B e antigen positive | 10052329 | |
| | | Hepatitis B reactivation | 10058827 | |
| | | Hepatitis B surface antigen | 10050529 | |
| | | Hepatitis B surface antigen positive | 10019742 | |
| | | Hepatitis B virus test | 10068415 | |
| | | Hepatitis B virus test positive | 10070217 | |
| | | Hepatitis A | 10019780 | |
| | | Hepatitis post | 10019791 | |
| | | transfusion | | |
| | | Hepatitis viral | 10019799 | |
| | | Withdrawal hepatitis | 10071220 | |
| Viral | HCV progression (V) | None | | Narrow |
| | | Chronic hepatitis C | 10008912 | Broad |
| | | Hepatitis C | 10019744 | |
| | | Hepatitis C RNA | 10019748 | |
| | | Hepatitis C RNA | 10068727 | |
| | | fluctuation | | |
| | | Hepatitis C RNA | 10068377 | |
| | | increased | | |
| | | Hepatitis C RNA | 10019750 | |
| | | positive | | |
| | | Hepatitis C virus test | 10068416 | |
| | | Hepatitis C virus test | 10070218 | |
| | Hornes simple: (IV) | positive Calitie harmas | 10051792 | Namer |
| | Herpes simplex (IV) | Colitis herpes | 10051782 | Narrow |
| | | Eczema herpeticum Gastritis harnes | 10014197 | |
| | | Gastritis herpes | 10051784 | |
| | | Herpes oesophagitis Herpes sepsis | 10052330<br>10058876 | |
| | | Herpes simplex colitis | 10038876 | _ |
| | | rierpes simplex confus | 100/4239 | |

| Category | Potential Opportunistic Infection | Preferred Term<br>(MedDRA Version<br>22.1) | Preferred Term<br>Code | Lilly Defined<br>Classification |
|---|---|---|---|---|
| | | Herpes simplex | 10019953 | |
| | | encephalitis | | |
| | | Herpes simplex gastritis | 10074240 | |
| | | Herpes simplex hepatitis | 10067389 | |
| | | Herpes simplex meningitis | 10019956 | |
| | | Herpes simplex meningoencephalitis | 10074247 | |
| | | Herpes simplex meningomyelitis | 10074250 | |
| | | Herpes simplex necrotising retinopathy | 10074252 | |
| | | Herpes simplex oesophagitis | 10074242 | |
| | | Herpes simplex pneumonia | 10065046 | |
| | | Herpes simplex sepsis | 10074246 | |
| | | Herpes simplex visceral | 10019963 | |
| | | Meningitis herpes | 10027242 | |
| | | Meningoencephalitis<br>herpetic | 10027285 | |
| | | Meningomyelitis herpes | 10074249 | |
| | | Pneumonia herpes viral | 10035703 | |
| | | Genital herpes simplex | 10073931 | |
| | | Herpes dermatitis | 10062639 | |
| | | Herpes pharyngitis | 10066888 | |
| | | Herpes simplex otitis externa | 10019959 | |
| | | Herpes simplex pharyngitis | 10074244 | |
| | | Ophthalmic herpes | 10073938 | |
| | | simplex | 10027700 | |
| | | Proctitis herpes Kaposi's varicelliform | 10036780<br>10051891 | |
| | | eruption Herpes simplex test | 10077969 | Broad |
| | | positive | | |
| | | Herpes simplex | 10019948 | _ |
| | | Herpes virus infection | 10019973 | _ |
| | | Nasal herpes | 10074936 | _ |
| | | Oral herpes | 10067152 | _ |
| | Herpes zoster (any | Genital herpes Disseminated varicella | 10018150<br>10076667 | Narrow |
| | form) (II) | zoster vaccine virus infection | 100/000/ | Ivaiiow |

| Category | Potential Opportunistic Infection | Preferred Term<br>(MedDRA Version<br>22.1) | Preferred Term<br>Code | Lilly Defined<br>Classification |
|---|---|---|---|---|
| | Infection | Encephalitis post | 10014603 | |
| | | varicella | 10014003 | |
| | | Genital herpes zoster | 10072210 | |
| | | Herpes zoster | 10019974 | |
| | | Herpes zoster cutaneous | 10074297 | |
| | | disseminated | 1007 1257 | |
| | | Herpes zoster | 10065038 | |
| | | disseminated | | |
| | | Herpes zoster infection | 10061208 | |
| | | neurological | | |
| | | Herpes zoster meningitis | 10074259 | |
| | | Herpes zoster | 10074248 | |
| | | meningoencephalitis | | |
| | | Herpes zoster | 10074251 | |
| | | meningomyelitis | | |
| | | Herpes zoster | 10079327 | |
| | | meningoradiculitis | | |
| | | Herpes zosternecrotising | 10074253 | |
| | | retinopathy | | |
| | | Herpes zoster oticus | 10063491 | |
| | | Herpes zoster | 10074245 | |
| | | pharyngitis | | |
| | | Necrotising herpetic | 10065119 | |
| | | retinopathy | | |
| | | Ophthalmic herpes | 10030865 | |
| | | zoster | | |
| | | Varicella | 10046980 | |
| | | Varicella keratitis | 10077496 | |
| | | Varicella post vaccine | 10063522 | |
| | | Varicella zoster gastritis | 10074241 | |
| | | Varicella zoster | 10074243 | |
| | | oesophagitis | | |
| | | Varicella zoster | 10074254 | |
| | | pneumonia | | |
| | | Varicella zoster virus | 10075611 | |
| | | infection | | |
| | | Herpes ophthalmic | 10062004 | |
| | | Varicella virus test | 10070444 | Broad |
| | | Varicella virus test | 10070214 | |
| | | positive | 10055101 | ) T |
| | | BK virus infection | 10055181 | Narrow |
| | | Human polyomavirus | 10057366 | |
| | | infection | 10074261 | _ |
| | | JC virus granule cell | 10074361 | |
| | | neuronopathy | | |

| Category | Potential<br>Opportunistic<br>Infection | Preferred Term<br>(MedDRA Version<br>22.1) | Preferred Term<br>Code | Lilly Defined<br>Classification |
|---|---|---|---|---|
| | II D 1 | JC virus infection | 10023163 | |
| | Human Polyomavirus infection including | Polyomavirus-associated nephropathy | 10065381 | |
| | BK virus disease and PVAN (V), and | Progressive multifocal leukoencephalopathy | 10036807 | |
| | Progressive<br>Multifocal | JC virus test | 10068794 | Broad |
| | Leukoencephalopathy | Polyomavirus test | 10075038 | |
| | (IV) | Polyomavirus test positive | 10070342 | |
| | Post-transplant<br>lymphoproliferative<br>disorder (EBV) (V) | Epstein-Barr virus associated lymphoproliferative | 10068349 | Narrow |
| | | disorder Post transplant lymphoproliferative disorder | 10051358 | |
| | | Epstein-Barr viraemia | 10065110 | Broad |
| | | Epstein-Barr virus associated lymphoma | 10071441 | |
| | | Epstein-Barr virus infection | 10015108 | |
| | | Lymphoproliferative disorder | 10061232 | |
| | | Lymphoproliferative disorder in remission | 10061233 | |
| | | Oral hairy leukoplakia | 10030979 | |
| Parasites | Trypanosoma cruzi | None | | Narrow |
| | infection (Chagas' Disease) | American trypanosomiasis | 10001935 | Broad |
| | (disseminated disease | Trypanosomiasis | 10044707 | |
| | only) (V) | Meningitis<br>trypanosomal | 10027258 | |
| | Cryptosporidium species (chronic | Biliary tract infection cryptosporidial | 10067319 | Narrow |
| | disease only) (IV) | Cryptosporidiosis infection | 10011502 | Broad |
| | | Gastroenteritis cryptosporidial | 10017899 | |
| | Leishmaniasis | Visceral leishmaniasis | 10047505 | Narrow |
| | (Visceral only) (IV) | Leishmaniasis | 10024198 | Broad |
| | Stronglyoides<br>(hyperinfection | None | 13021170 | Narrow |
| | syndrome and<br>disseminated forms<br>only) (IV) | Strongyloidiasis | 10042254 | Broad |

| Category | Potential Opportunistic Infection | Preferred Term<br>(MedDRA Version<br>22.1) | Preferred Term<br>Code | Lilly Defined<br>Classification |
|---|---|---|---|---|
| | Toxoplasmosis (IV) | Cerebral toxoplasmosis | 10057854 | Narrow |
| | | Eye infection | 10015939 | |
| | | toxoplasmal | | |
| | | Hepatitis toxoplasmal | 10019798 | |
| | | Meningitis toxoplasmal | 10048848 | |
| | | Myocarditis toxoplasmal | 10028617 | |
| | | Pneumonia toxoplasmal | 10067566 | |
| | | Toxoplasma serology | 10050941 | Broad |
| | | Toxoplasmosis | 10044272 | |
| Non-specific | Non-specific terms | None | | Narrow |
| terms | 1 | Delftia acidovorans | 10081339 | |
| | | infection | | |
| | | Sphingomonas | 10081563 | |
| | | paucimobilis | | |
| | | bacteraemia | | |
| | | Central nervous system | | Broad |
| | | immune reconstitution | 10080100 | |
| | | inflammatory response | | |
| | | Abscess fungal | 10000269 | |
| | | Alternaria infection | 10054207 | |
| | | Arthritis fungal | 10060966 | |
| | | Biliary tract infection | 10065203 | |
| | | fungal | | |
| | | Central nervous system | 10072805 | |
| | | fungal infection | | |
| | | Cerebral fungal | 10049657 | |
| | | infection | | |
| | | Encephalitis fungal | 10065170 | |
| | | Erythema induratum | 10015213 | |
| | | Eye infection fungal | 10015933 | |
| | | Fungaemia | 10017523 | |
| | | Fungal abscess central | 10017524 | |
| | | nervous system | | |
| | | Fungal endocarditis | 10017529 | |
| | | Fungal labyrinthitis | 10065174 | |
| | | Fungal oesophagitis | 10049656 | |
| | | Fungal peritonitis | 10061138 | |
| | | Fungal pharyngitis | 10076516 | |
| | | Fungal retinitis | 10068613 | |
| | | Fungal sepsis | 10058872 | |
| | | Fungal urethritis | 10081163 | |
| | | Hepatic infection fungal | 10065217 | |
| | | Meningitis fungal | 10027236 | |
| | | Mycotic | 10063202 | |
| | | endophthalmitis | | |

| Category | Potential Opportunistic Infection | Preferred Term<br>(MedDRA Version<br>22.1) | Preferred Term<br>Code | Lilly Defined<br>Classification |
|---|---|---|---|---|
| | Infection | , | 10050026 | |
| | | Myocarditis mycotic | 10059026 | - |
| | | Oral fungal infection | 10061324 | |
| | | Oropharyngitis fungal | 10061891 | |
| | | Osteomyelitis fungal | 10065239 | |
| | | Otitis media fungal | 10065175 | |
| | | Pancreatitis fungal | 10065190 | |
| | | Pericarditis fungal | 10065220 | |
| | | Phaehyphomycosis | 10034799 | |
| | | Pneumonia fungal | 10061354 | |
| | | Pulmonary mycosis | 10037422 | |
| | | Pulmonary | 10068184 | |
| | | trichosporonosis | | |
| | | Sinusitis fungal | 10058678 | |
| | | Splenic infection fungal | 10065194 | |
| | | Systemic mycosis | 10052366 | |
| Pneumonia | Infective Pneumonia SMQ | All PTs | 20000231 | Narrow |

Abbreviations: DNA = deoxyribonucleic acid; EBV= Epstein-Barr virus; HBV = hepatitis B virus; MedDRA = Medical Dictionary for Regulatory Activities; PT = preferred term; PVAN = Polyomavirus-associated nephropathy; SMQ = standardized MedDRA query.

6.9. Appendix 9: List of MedDRA Preferred Terms for Elevated or Increased Lipids from the Dyslipidemia SMQ (SMQ20000026)

| Preferred Term (MedDRA Version 20.0) | Preferred Term Code |
|-----------------------------------------------------|---------------------|
| Apolipoprotein B/Apolipoprotein A-1 ratio increased | 10065516 |
| Autoimmune hyperlipidaemia | 10071577 |
| Blood cholesterol abnormal | 10005423 |
| Blood cholesterol increased | 10005425 |
| Blood triglycerides abnormal | 10005837 |
| Blood triglycerides increased | 10005839 |
| Diabetic dyslipidaemia | 10070901 |
| Dyslipidaemia | 10058108 |
| Familial hypertriglyceridaemia | 10059183 |
| Fat overload syndrome | 10074028 |
| High density lipoprotein abnormal | 10020051 |
| High density lipoprotein decreased | 10020060 |
| High density lipoprotein increased | 10020061 |
| Hypercholesterolaemia | 10020603 |
| Hyperlipidaemia | 10062060 |
| Hypertriglyceridaemia | 10020869 |
| Hypo HDL cholesterolaemia | 10068961 |

| Intermediate density lipoprotein increased | 10064236 |
|----------------------------------------------------|----------|
| LDL/HDL ratio increased | 10049030 |
| Lipid metabolism disorder | 10061227 |
| Lipids abnormal | 10024588 |
| Lipids increased | 10024592 |
| Lipoprotein (a) abnormal | 10054023 |
| Lipoprotein (a) increased | 10054009 |
| Low density lipoprotein abnormal | 10024901 |
| Low density lipoprotein increased | 10024910 |
| Non-high-density lipoprotein cholesterol increased | 10063967 |
| Remnant hyperlipidaemia | 10038316 |
| Total cholesterol/HDL ratio abnormal | 10058633 |
| Total cholesterol/HDL ratio increased | 10058630 |
| Type I hyperlipidaemia | 10060749 |
| Type II hyperlipidaemia | 10045254 |
| Type IIa hyperlipidaemia | 10045261 |
| Type IIb hyperlipidaemia | 10045263 |
| Type III hyperlipidaemia | 10060751 |
| Type IV hyperlipidaemia | 10060753 |
| Type V hyperlipidaemia | 10060755 |
| Very low density lipoprotein abnormal | 10047352 |
| Very low density lipoprotein increased | 10047361 |

# 6.10. Appendix 10: List of Planned Laboratory Analytes with Reference Range Sources

| Laboratory | Laboratory Analyte | Reference | Analy | ysis Type |
|-------------|----------------------|------------|----------|---------------|
| Group/Order | | Range Name | Central | Outlier/Shift |
| | | | Tendency | Analysis |
| Hematology | | | | |
| 1 | Hemoglobin | LCTPB | Yes | Yes |
| 2 | Hematocrit | LCTPB | Yes | Yes |
| 3 | Erythrocyte Count | LCTPB | Yes | Yes |
| 4 | Mean Cell Volume | LCTPB | Yes | Yes |
| 5 | Mean Cell Hemoglobin | LCTPB | Yes | Yes |
| 6 | MCHC | LCTPB | Yes | Yes |
| 7 | Platelets | LCTPB | Yes | Yes |
| 8 | Leukocyte Count | LCTPB | Yes | Yes |
| 9 | Bands | LCTPB | Yes | Yes |
| 10 | Neutrophils | LCTPB | Yes | Yes |
| 11 | Lymphocytes | LCTPB | Yes | Yes |
| 12 | Monocytes | LCTPB | Yes | Yes |
| 13 | Eosinophils | LCTPB | Yes | Yes |
| 14 | Basophils | LCTPB | Yes | Yes |

| Laboratory<br>Group/Order | Laboratory Analyte | Reference<br>Range Name | Analysis Type | |
|---|---|---|---|---|
| | | | Central<br>Tendency | Outlier/Shift<br>Analysis |
| 1 | ALT/SGPT | Labcorp | Yes | Yes |
| 2 | AST/SGOT | Labcorp | Yes | Yes |
| 3 | Alkaline Phosphatase | Labcorp | Yes | Yes |
| 4 | Total Bilirubin | Labcorp | Yes | Yes |
| 5 | Direct Bilirubin | Labcorp | Yes | Yes |
| 6 | Albumin | LCTPB | Yes | Yes |
| 7 | Creatine Phosphokinase | LCTPB | Yes | Yes |
| 8 | Creatinine | Labcorp | Yes | Yes |
| 9 | Urea Nitrogen | LCTPB | Yes | Yes |
| 11 | estimated GFR | Labcorp | Yes | Yes |
| 12 | Creatinine Clearance | Labcorp | Yes | Yes |
| 13 | Sodium | LCTPB | Yes | Yes |
| 14 | Potassium | LCTPB | Yes | Yes |
| 15 | Calcium | LCTPB | Yes | Yes |
| 16 | Total Protein | LCTPB | Yes | Yes |
| 17 | Fasting Glucose | LCTPB | Yes | Yes |
| 18 | Glucose, Non-Fasting or Random | LCTPB | Yes | Yes |
| 19 | Uric Acid | LCTPB | Yes | Yes |
| 20 | Cholesterol | LCTPB | Yes | Yes |
| 21 | Triglycerides | LCTPB | Yes | Yes |
| 22 | LDL Cholesterol – Direct | Labcorp | Yes | Yes |
| 23 | HDL Cholesterol – Direct | Labcorp | Yes | Yes |
| 24 | LDL/HDL Ratio - Calculated | None | Yes | No |
| Immunoglobu | lins | | | |
| 1 | Immunoglobulin A | Labcorp | Yes | Yes |
| 2 | Immunoglobulin G | Labcorp | Yes | Yes |
| 3 | Immunoglobulin M | Labcorp | Yes | Yes |
| Urinalysis | | | | |
| 1 | Specific Gravity | LCTPB | Yes | Yes |
| 2 | pН | LCTPB | Yes | Yes |
| 3 | UA-color | None | No | Yes |
| 4 | UA-glucose | None | No | Yes |
| 5 | UA-protein | None | No | Yes |
| 6 | UA-bilirubin | None | No | Yes |
| 7 | UA-urobilinogen | None | No | Yes |
| 8 | UA-nitrites | None | No | Yes |
| 9 | UA-leukoesterase | None | No | Yes |
| 10 | UA-ketones | None | No | Yes |
| 11 | UA-occult blood | None | No | Yes |
| Flow Cytomet | | | | |
| 1 | CD3+ T Cells – % | Labcorp | Yes | Yes |
| 2 | CD3+ T Cells – Absolute | Labcorp | Yes | Yes |
| 3 | CD3+CD4+ T cells (CD4) – % | Labcorp | Yes | Yes |
| J | | | | |
| 4 | CD3+CD4+ T cells (CD4) – Absolute | Labcorp | Yes | Yes |

| Laboratory<br>Group/Order | Laboratory Analyte | Reference<br>Range Name | Analy | ysis Type |
|---|---|---|---|---|
| | | | Central | Outlier/Shift |
| | | | Tendency | Analysis |
| 6 | CD3+CD8+ T cells (CD8) – Absolute | Labcorp | Yes | Yes |
| 7 | CD56+/CD16+ NK cells - % | Labcorp | Yes | Yes |
| 8 | CD56+/CD16+ NK cells – Absolute | Labcorp | Yes | Yes |
| ) | CD19+ B cells – % | Labcorp | Yes | Yes |
| 10 | CD19+ B cells – Absolute | Labcorp | Yes | Yes |
| 11 | CD4+CXCR3+CCR6- Th1 cells - % | None | Yes | No |
| 12 | CD4+CXCR3+CCR6- Th1 cells - Absolute | None | Yes | No |
| 13 | CD4+CXCR3-CCR6+ Th17 cells - % | None | Yes | No |
| 14 | CD4+CXCR3-CCR6+ Th17 cells - Absolute | None | Yes | No |
| 15 | CD3+CD4+CD127-<br>/loCD25+FoxP3+ (CD4+) T<br>regulatory cells - % | None | Yes | No |
| 16 | CD3+CD4+CD127-<br>/loCD25+FoxP3+ (CD4+) T<br>regulatory cells - Absolute | None | Yes | No |
| 17 | CD3+CD4+CD127-/loCD25+<br>(CD4+) IL2-producing naïve and<br>central memory Helper T cells - % | None | Yes | No |
| 18 | CD3+CD4+CD127-/loCD25+<br>(CD4+) IL2-producing naïve and<br>central memory Helper T cells -<br>Absolute | None | Yes | No |
| 19 | CD20+ B cells – % | None | Yes | No |
| 20 | CD20+ B cells – Absolute | None | Yes | No |
| 21 | CD19+CD27-IgD+ mature naïve B cells – % | None | Yes | No |
| 22 | CD19+CD27-IgD+ mature naïve B cells – Absolute | None | Yes | No |
| 23 | CD19+CD27+IgD- switched memory B cells – % | None | Yes | No |
| 24 | CD19+CD27+IgD- switched memory B – Absolute | None | Yes | No |
| 25 | CD19+CD27+IgD+ non-switched memory B cells – % | None | Yes | No |
| 26 | CD19+CD27+IgD+ non-switched memory B – Absolute | None | Yes | No |
| 27 | CD19+CD27-IgD-<br>Immature/transitional B cells – % | None | Yes | No |
| 28 | CD19+CD27-IgD-<br>Immature/transitional B – Absolute | None | Yes | No |
| 29 | CD4/CD8 Ratio - Calculated | None | Yes | No |
| | CD4+CD45RA-CCR7- effector memory T cells | None | No | No |

| Laboratory | boratory Laboratory Analyte Reference | Reference | Analysis Type | |
|---|---|---|---|---|
| Group/Order | | Range Name | Central<br>Tendency | Outlier/Shift<br>Analysis |
| | CD4+CD45RA+CCR7- effector memory T cells | None | No | No |
| | CD4+CD45RA+CCR7- naïve T cells | None | No | No |
| | CD4+CD45RA-CCR7+ central memory T cells | None | No | No |
| | CD8+CD45RA+CCR7+ naïve T cells | None | No | No |
| | CD8+CD45RA-CCR7+ central memory T cells | None | No | No |
| | CD8+CD45RA-CCR7- effector<br>memory T cells | None | No | No |
| | CD8+CD45RA+CCR7- effector memory T cells | None | No | No |

Abbreviations: ALT/SGPT = alanine aminotransferase/serum glutamic pyruvic transaminase; AST/SGOT = aspartate aminotransferase/serum glutamic oxaloacetic transaminase; CD = cluster of differentiation; eGFR = estimated glomerular filtration rate; HDL = high-density lipoprotein; LCTPB = Lilly Large Clinical Trial Population Based; LDL = low-density lipoprotein; MCHC = mean corpuscular hemoglobin concentration; NK = natural killer; UA = urinalysis.

## 7. References

- Bretz F, Pinheiro JC, Branson M. Combining multiple comparisons and modeling techniques in dose-response studies. Biometrics. 2005;61(3):738-748. https://doi.org/ 10.1111/j.1541-0420.2005.00344.x
- [FDA] Food and Drug Administration. E9(R1): statistical principles for clinical trials: addendum: estimands and sensitivity analyses in clinical trials: guidance for industry. Draft Guidance. Available at:
  - https://www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidance s/UCM582738.pdf. Published 16 June 2017. Accessed 23 November 2019.
- [FDA] Food and Drug Administration. Qualification of the MCP-Mod Procedure. Available at: FDA Qualification of MCP-MOD Method. Application date 22 April 2015.
- Gould AL. BMA-Mod: A Bayesian model averaging strategy for determining dose-response relationships in the presence of model uncertainty. Biom J. 2019;61(5):1141-1159. https://doi.org/ 10.1002/bimj.201700211

# Signature Page for VV-CLIN-023696 v1.0

| Approval | PPD |
|----------|-------------------------------|
| | Statistician |
| | 18-Mar-2022 02:51:35 GMT+0000 |

Signature Page for VV-CLIN-023696 v1.0